CLINICAL TRIAL: NCT03091920
Title: A Phase 2 Study to Compare the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of 2 Dose Regimens of IW-1973 in Patients With Stable Type 2 Diabetes and Hypertension
Brief Title: Trial of IW-1973, A Stimulator of Soluble Guanylate Cyclase (sGC) in Patients With Stable Type 2 Diabetes and Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cyclerion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C1973-202
Record Dates: First submitted 2017-03-08; First posted 2017-03-27 (Actual); Results first posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — praliciguat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IW-1973 QD/QD (Experimental): On Days 1-14: IW-1973 40 mg taken once daily (QD) in morning (AM) and placebo taken QD at night (PM).
  Interventions: Drug: IW-1973; Drug: Placebo
- IW-1973 BID (Twice Daily)/QD (Experimental): On Days 1-7: IW-1973 20 mg taken in AM and IW-1973 20 mg taken in PM. On Days 8-14: IW-1973 40 mg taken QD in AM and placebo taken QD in PM.
  Interventions: Drug: IW-1973; Drug: Placebo
- Placebo (Placebo Comparator): On Days 1-14: Placebo taken in AM and in PM.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IW-1973 — Oral Tablet
  Arms: IW-1973 BID (Twice Daily)/QD; IW-1973 QD/QD
Drug: Placebo — Oral Tablet

SUMMARY:
To compare the safety, tolerability, pharmacokinetic (PK) profile, and pharmacodynamic (PD) effects of 2 treatment regimens of IW-1973 tablet (40 mg per day) administered orally for 2 weeks to patients with stable type 2 diabetes mellitus and hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ambulatory male or female
* Patient's body mass index score is > 20 and < 40 kg/m^2 at the Screening Visit
* Women of childbearing potential must have a negative pregnancy test at the time of screening and check-in and must agree to use protocol-specified contraception throughout the duration of the study
* Patient's health is stable with no clinically significant findings on physical examination
* Patient has type 2 (ie, adult onset) diabetes mellitus diagnosed by a physician or nurse practitioner > 6 months before the Screening Visit, is on a stable glycemic control medication, and protocol specified hemoglobin (Hb)A1c values at the Screening Visit
* Patient has hypertension diagnosed by a physician or nurse practitioner > 6 months before the Screening Visit, and blood pressure (BP) within the protocol's acceptable range
* Patients must be on a stable regimen for hypertension control that includes an angiotensin converting enzyme inhibitor (ACEi) or angiotensin receptor blocker (ARB), stable for 28 days
* Other inclusion criteria per protocol

Exclusion Criteria:

* Patient has a clinically significant active or unstable medical condition that, in the opinion of the Investigator, would preclude trial participation
* Patient is on medication(s) that, when co-administered with a sGC stimulator, could increase the risk of hypotension
* Patient has evidence of severe or active end-organ damage
* Patient is an active smoker or has used any nicotine-containing products (cigarettes, e-cigarettes, vape pens, cigars, chewing tobacco, gum, patches) during the 6 months before Check-in. Use of nicotine is excluded during the study until after the End of Trial Visit.
* Other exclusion criteria per protocol

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2017-08-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ProSciento, Inc., Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hanrahan JP, Seferovic JP, Wakefield JD, Wilson PJ, Chickering JG, Jung J, Carlson KE, Zimmer DP, Frelinger AL 3rd, Michelson AD, Morrow L, Hall M, Currie MG, Milne GT, Profy AT. An exploratory, randomised, placebo-controlled, 14 day trial of the soluble guanylate cyclase stimulator praliciguat in participants with type 2 diabetes and hypertension. Diabetologia. 2020 Apr;63(4):733-743. doi: 10.1007/s00125-019-05062-x. Epub 2019 Dec 19. PMID 31858186

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo oral tablet taken morning (AM) and night (PM) on Days 1-14.
- IW-1973 40 mg Twice Dily (BID)/Once Daily (QD): IW-1973 20 mg oral tablet taken in AM and 20 mg oral tablet taken in PM on Days 1-7.
  IW-1973 40 mg oral tablet taken QD in AM and placebo oral tablet taken QD in PM on Days 8-14.
- IW-1973 40 mg QD/QD: IW-1973 40 mg oral tablet taken QD in AM and placebo taken QD in PM on Days 1-14.
Period: Overall Study
Arm/Group | Placebo | IW-1973 40 mg Twice Dily (BID)/Once Daily (QD) | IW-1973 40 mg QD/QD
Started | 6 | 10 | 10
Completed | 6 | 9 | 10
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo oral tablet taken in AM and in PM on Days 1-14.
- IW-1973 40 mg BID/QD: IW-1973 20 mg oral tablet taken in AM and 20 mg oral tablet taken in PM on Days 1-7.
  IW-1973 40 mg oral tablet taken QD in AM and placebo oral tablet taken QD in PM on Days 8-14.
- Total: Total of all reporting groups
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD | Total
Number analyzed (Participants) | 6 | 10 | 10 | 26
Age, Customized [Count of Participants; unit: Participants]
  40 to < 65 years old | 4 | 6 | 7 | 17
  >= 65 years old | 2 | 4 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 5 | 13
  Male | 2 | 6 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 3 | 10
  Not Hispanic or Latino | 1 | 8 | 7 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 7 | 7 | 20
  Asian | 0 | 1 | 2 | 3
  Black or African American | 0 | 2 | 1 | 3
Percentage of Participants With Baseline Supine BP Less Than 130/80 mmHg [Number; unit: percentage of participants] | 33.3 | 80.0 | 60.0 | 70.0

OUTCOME MEASURES:

1. Primary Outcome: Change From Study Baseline Over Time in Supine Systolic Blood Pressure
Time Frame: Study Baseline (Day 1 predose AM); Days 2-14: predose AM; Days 1, 2, 7, 8, 13: postdose AM 1 hour and 4 hour; Day 1: postdose AM 8 hour; Days 1, 2, 8, 13: predose PM; Days 1, 2: postdose PM 1 hour; Days 2, 3: postdose PM 4 hour; Days 15, 21, 42
Population: Pharmacodynamic (PD) Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
mmHg
  Study Baseline (Day 1 predose AM) | 130.2 (11.1) | 120.1 (8.9) | 128.6 (10.1)
  Day 1 postdose AM: 1 hour | -6.8 (4.8) | -7.7 (3.9) | -6.2 (3.7)
  Day 1 postdose AM: 4 hour | 4.4 (6.0) | -9.5 (4.9) | -11.1 (4.6)
  Day 1 postdose AM: 8 hour | 0.5 (5.0) | -9.4 (4.0) | -2.7 (3.8)
  Day 1 predose PM | 1.8 (6.3) | -6.9 (5.1) | -1.7 (4.8)
  Day 1 postdose PM: 1 hour | -0.6 (5.6) | -3.9 (4.5) | -5.0 (4.3)
  Day 2 predose AM | 5.5 (3.5) | -2.9 (2.8) | -0.2 (2.7)
  Day 2 postdose AM: 1 hour | 2.0 (4.6) | -13.4 (3.7) | -7.4 (3.5)
  Day 2 postdose AM: 4 hour | 1.7 (6.1) | -7.1 (4.9) | -9.4 (4.7)
  Day 2 predose PM | 4.6 (4.5) | -7.1 (3.6) | -2.4 (3.4)
  Day 2 postdose PM: 1 hour | -3.8 (5.3) | -2.2 (4.3) | -3.1 (4.1)
  Day 2 postdose PM: 4 hour | -5.0 (4.2) | -9.7 (3.4) | -8.0 (3.3)
  Day 3 predose AM | -0.8 (4.0) | -5.5 (3.2) | -6.5 (3.1)
  Day 3 postdose PM: 4 hour | -5.8 (4.8) | -6.0 (3.9) | -8.6 (3.7)
  Day 4 predose AM | -0.8 (3.3) | -7.0 (2.7) | -8.9 (2.6)
  Day 5 predose AM | -0.2 (3.6) | -1.9 (2.9) | -10.3 (2.8)
  Day 6 predose AM | -4.3 (4.1) | -11.0 (3.3) | -8.6 (3.2)
  Day 7 predose AM | -4.3 (4.8) | -3.3 (3.8) | -8.1 (3.7)
  Day 7 postdose AM: 1 hour | -5.3 (4.4) | -8.4 (3.5) | -11.7 (3.4)
  Day 7 postdose AM: 4 hour | 1.3 (4.8) | -8.2 (3.9) | -15.9 (3.7)
  Day 8 predose AM | 3.7 (4.6) | -8.0 (3.7) | -4.7 (3.6)
  Day 8 postdose AM: 1 hour | -2.0 (5.3) | -15.4 (4.3) | -12.3 (4.1)
  Day 8 postdose AM: 4 hour | -5.2 (6.1) | -15.2 (4.9) | -9.8 (4.7)
  Day 8 predose PM | -4.5 (5.5) | -8.8 (4.4) | -5.8 (4.2)
  Day 9 predose AM | 3.0 (3.7) | -9.7 (3.0) | -2.1 (2.9)
  Day 10 predose AM | -1.3 (4.0) | -9.3 (3.2) | -5.1 (3.0)
  Day 11 predose AM | 3.8 (5.4) | -12.3 (4.4) | -4.5 (4.2)
  Day 12 predose AM | -6.5 (4.1) | -9.8 (3.3) | -12.0 (3.1)
  Day 13 predose AM | -1.6 (3.7) | -13.5 (3.0) | -8.1 (2.8)
  Day 13 postdose AM: 1 hour | -2.4 (4.0) | -16.6 (3.2) | -14.2 (3.1)
  Day 13 postdose AM: 4 hour | -3.9 (6.3) | -15.6 (5.1) | -13.7 (4.8)
  Day 13 predose PM | -1.9 (4.0) | -13.2 (3.2) | -11.8 (3.1)
  Day 14 predose AM | -3.7 (5.9) | -9.5 (4.7) | -9.8 (4.5)
  Day 15/Discharge | 2.1 (4.9) | -6.0 (4.0) | -3.0 (3.8)
  Day 21/Follow-Up | -3.5 (4.3) | 1.3 (3.5) | 1.7 (3.3)
  Day 42/End of Trial | 3.3 (6.2) | 8.8 (5.0) | -1.2 (4.8)
Statistical Analysis 1: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1 postdose AM 1 hour; Test type: Other — No statistical testing was performed; LS Mean Difference = -0.9, 95% CI 2-sided [-14.2 to 12.4], Standard Error of Mean 6.4 — LS mean difference and associated 95% confidence interval (CI) is from an analysis of covariance (ANCOVA) model with treatment as fixed effect and baseline as covariate. Standard Error of the Mean=Standard Error of the LS Mean Difference
Statistical Analysis 2: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1 postdose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.6, 95% CI 2-sided [-11.8 to 12.9], Standard Error of Mean 6.0 — Least Squares mean difference and associated 95% CI is from an ANCOVA model with treatment as fixed effect and baseline as covariate
Statistical Analysis 3: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1 postdose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -13.9, 95% CI 2-sided [-30.6 to 2.8], Standard Error of Mean 8.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1 postdose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -15.5, 95% CI 2-sided [-31.0 to 0], Standard Error of Mean 7.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1 postdose AM 8 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -9.9, 95% CI 2-sided [-23.8 to 3.9], Standard Error of Mean 6.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1 postdose AM 8 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.1, 95% CI 2-sided [-16.0 to 9.7], Standard Error of Mean 6.2 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1 predose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = -8.8, 95% CI 2-sided [-26.2 to 8.6], Standard Error of Mean 8.4 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1 predose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.6, 95% CI 2-sided [-19.7 to 12.6], Standard Error of Mean 7.8 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1 postdose PM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.3, 95% CI 2-sided [-18.7 to 12.2], Standard Error of Mean 7.5
Statistical Analysis 10: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1 postdose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.4, 95% CI 2-sided [-18.7 to 9.9], Standard Error of Mean 6.9 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 2 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -8.5, 95% CI 2-sided [-18.2 to 1.3], Standard Error of Mean 4.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 12: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 2 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.7, 95% CI 2-sided [-14.8 to 3.3], Standard Error of Mean 4.4 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 2 postdose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -15.4, 95% CI 2-sided [-28.1 to -2.8], Standard Error of Mean 6.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 14: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 2 postdose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -9.4, 95% CI 2-sided [-21.1 to 2.3], Standard Error of Mean 5.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 2 postdose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -8.8, 95% CI 2-sided [-25.6 to 7.9], Standard Error of Mean 8.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 16: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 2 postdose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -11.2, 95% CI 2-sided [-26.7 to 4.4], Standard Error of Mean 7.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 2 predose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = -11.7, 95% CI 2-sided [-24.0 to 0.6], Standard Error of Mean 5.9 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 18: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 2 predose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = -7.0, 95% CI 2-sided [-18.4 to 4.4], Standard Error of Mean 5.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 2 postdose PM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.6, 95% CI 2-sided [-13.0 to 16.2], Standard Error of Mean 7.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 20: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 2 postdose PM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.7, 95% CI 2-sided [-12.9 to 14.2], Standard Error of Mean 6.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 2 postdose PM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.7, 95% CI 2-sided [-16.4 to 7.1], Standard Error of Mean 5.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 22: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 2 postdose PM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.0, 95% CI 2-sided [-13.9 to 7.9], Standard Error of Mean 5.2 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 3 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.7, 95% CI 2-sided [-15.8 to 6.4], Standard Error of Mean 5.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 24: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 3 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.8, 95% CI 2-sided [-16.0 to 4.5], Standard Error of Mean 5.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 25: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 3 postdose PM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.2, 95% CI 2-sided [-13.6 to 13.1], Standard Error of Mean 6.4 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 26: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 3 postdose PM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.8, 95% CI 2-sided [-15.2 to 9.6], Standard Error of Mean 6.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 27: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 4 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -6.2, 95% CI 2-sided [-15.5 to 3.0], Standard Error of Mean 4.4 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 28: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 4 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -8.1, 95% CI 2-sided [-16.6 to 0.5], Standard Error of Mean 4.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 29: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 5 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.7, 95% CI 2-sided [-11.8 to 8.4], Standard Error of Mean 4.9 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 30: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 5 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -10.0, 95% CI 2-sided [-19.4 to -0.7], Standard Error of Mean 4.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 31: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 6 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -6.7, 95% CI 2-sided [-18.1 to 4.7], Standard Error of Mean 5.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 32: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 6 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.3, 95% CI 2-sided [-14.8 to 6.3], Standard Error of Mean 5.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 33: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.0, 95% CI 2-sided [-12.2 to 14.1], Standard Error of Mean 6.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 34: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.8, 95% CI 2-sided [-16.0 to 8.4], Standard Error of Mean 5.9 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 35: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7 postdose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.0, 95% CI 2-sided [-15.1 to 9.1], Standard Error of Mean 5.8 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 36: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7 postdose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -6.4, 95% CI 2-sided [-17.6 to 4.8], Standard Error of Mean 5.4 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 37: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7 postdose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -9.5, 95% CI 2-sided [-22.7 to 3.7], Standard Error of Mean 6.4 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 38: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7 postdose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -17.2, 95% CI 2-sided [-29.5 to -5.0], Standard Error of Mean 5.9 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 39: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 8 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -11.7, 95% CI 2-sided [-24.4 to 1.1], Standard Error of Mean 6.2 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 40: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 8 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -8.3, 95% CI 2-sided [-20.2 to 3.5], Standard Error of Mean 5.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 41: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 8 postdose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -13.4, 95% CI 2-sided [-28.1 to 1.4], Standard Error of Mean 7.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 42: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 8 postdose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -10.3, 95% CI 2-sided [-24.0 to 3.3], Standard Error of Mean 6.6 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 43: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 8 postdose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -10.1, 95% CI 2-sided [-27.0 to 6.9], Standard Error of Mean 8.2 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 44: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 8 postdose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.6, 95% CI 2-sided [-20.4 to 11.1], Standard Error of Mean 7.6 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 45: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 8 predose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.2, 95% CI 2-sided [-19.5 to 11.0], Standard Error of Mean 7.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 46: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 8 predose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.3, 95% CI 2-sided [-15.4 to 12.8], Standard Error of Mean 6.8 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 47: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 9 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -12.7, 95% CI 2-sided [-23.0 to -2.5], Standard Error of Mean 5.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 48: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 9 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.2, 95% CI 2-sided [-14.7 to 4.3], Standard Error of Mean 4.6 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 49: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 10 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -8.0, 95% CI 2-sided [-19.0 to 2.9], Standard Error of Mean 5.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 50: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 10 predose; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.8, 95% CI 2-sided [-14.0 to 6.3], Standard Error of Mean 4.9 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 51: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 11 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -16.1, 95% CI 2-sided [-31.0 to -1.2], Standard Error of Mean 7.2 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 52: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 11 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -8.3, 95% CI 2-sided [-22.1 to 5.6], Standard Error of Mean 6.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 53: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 12 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.4, 95% CI 2-sided [-14.6 to 7.9], Standard Error of Mean 5.4 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 54: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 12 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.5, 95% CI 2-sided [-15.9 to 4.9], Standard Error of Mean 5.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 55: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 13 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -11.9, 95% CI 2-sided [-22.1 to -1.7], Standard Error of Mean 4.9 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 56: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 13 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -6.5, 95% CI 2-sided [-16.0 to 2.9], Standard Error of Mean 4.6 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 57: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 13 postdose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -14.3, 95% CI 2-sided [-25.4 to -3.2], Standard Error of Mean 5.4 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 58: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 13 postdose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -11.8, 95% CI 2-sided [-22.1 to -1.5], Standard Error of Mean 5.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 59: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 13 postdose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -11.7, 95% CI 2-sided [-29.0 to 5.6], Standard Error of Mean 8.4 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 60: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 13 postdose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -9.8, 95% CI 2-sided [-25.9 to 6.2], Standard Error of Mean 7.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 61: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 13 postdose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = -11.3, 95% CI 2-sided [-22.4 to -0.1], Standard Error of Mean 5.4 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 62: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 13 predose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = -9.9, 95% CI 2-sided [-20.2 to 0.4], Standard Error of Mean 5.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 63: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.8, 95% CI 2-sided [-22.0 to 10.5], Standard Error of Mean 7.8 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 64: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14 predose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -6.1, 95% CI 2-sided [-21.1 to 9.0], Standard Error of Mean 7.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 65: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 15 / Discharge; Test type: Other — No statistical testing was performed; Least squares mean difference = -8.1, 95% CI 2-sided [-21.7 to 5.6], Standard Error of Mean 6.6 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 66: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 15 / Discharge; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.0, 95% CI 2-sided [-17.7 to 7.6], Standard Error of Mean 6.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 67: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 21 / Follow-up; Test type: Other — No statistical testing was performed; Least squares mean difference = 4.8, 95% CI 2-sided [-7.0 to 16.7], Standard Error of Mean 5.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 68: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 21 / Follow-up; Test type: Other — No statistical testing was performed; Least squares mean difference = 5.2, 95% CI 2-sided [-5.8 to 16.2], Standard Error of Mean 5.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 69: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 42 / End of Trial; Test type: Other — No statistical testing was performed; Least squares mean difference = 5.5, 95% CI 2-sided [-11.7 to 22.6], Standard Error of Mean 8.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 70: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 42 / End of Trial; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.5, 95% CI 2-sided [-20.4 to 11.4], Standard Error of Mean 7.7 — [estimate comment as in outcome 1, analysis 2]

2. Primary Outcome: Change From Study Baseline Over Time in Supine Diastolic Blood Pressure
Time Frame: as for outcome 1
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
mmHg
  Study Baseline (Day 1 predose AM) | 80.3 (6.9) | 75.5 (4.4) | 74.8 (5.9)
  Day 1 postdose AM: 1 hour | -3.1 (2.4) | -5.7 (1.8) | -5.1 (1.8)
  Day 1 postdose AM: 4 hour | -0.3 (2.4) | -3.2 (1.8) | -7.4 (1.8)
  Day 1 postdose AM: 8 hour | 0.9 (2.3) | -4.6 (1.7) | -3.7 (1.7)
  Day 1 predose PM | -1.3 (2.2) | -4.9 (1.6) | -3.5 (1.6)
  Day 1 postdose PM: 1 hour | -0.9 (3.4) | -5.9 (2.5) | -3.7 (2.5)
  Day 2 predose AM | 3.1 (2.0) | -1.3 (1.5) | 0 (1.5)
  Day 2 postdose AM: 1 hour | -1.4 (2.4) | -8.1 (1.8) | -6.7 (1.8)
  Day 2 postdose AM: 4 hour | 2.2 (3.4) | -3.1 (2.5) | -6.2 (2.5)
  Day 2 predose PM | 1.9 (2.3) | -3.7 (1.7) | -2.6 (1.7)
  Day 2 postdose PM: 1 hour | -2.2 (2.6) | -2.7 (1.9) | -4.4 (1.9)
  Day 2 postdose PM: 4 hour | -3.9 (2.7) | -6.3 (2.0) | -5.4 (2.0)
  Day 3 predose AM | -0.8 (2.5) | -0.6 (1.8) | -0.5 (1.8)
  Day 3 postdose PM: 4 hour | -5.5 (3.0) | -4.0 (2.2) | -6.7 (2.2)
  Day 4 predose AM | 0.3 (2.2) | -4.0 (1.6) | -4.2 (1.6)
  Day 5 predose AM | 1.8 (2.2) | -0.6 (1.6) | -5.3 (1.6)
  Day 6 predose AM | -0.5 (1.9) | -3.3 (1.4) | -5.2 (1.4)
  Day 7 predose AM | 0.9 (2.9) | -3.2 (2.1) | -3.4 (2.1)
  Day 7 postdose AM: 1 hour | -1.7 (2.4) | -6.0 (1.8) | -7.4 (1.8)
  Day 7 postdose AM: 4 hour | -6.1 (3.5) | -5.1 (2.6) | -5.9 (2.6)
  Day 8 predose AM | 0.6 (2.7) | -3.9 (1.9) | -2.2 (2.0)
  Day 8 postdose AM: 1 hour | 0 (2.4) | -9.3 (1.8) | -8.3 (1.8)
  Day 8 postdose AM: 4 hour | -3.6 (2.8) | -8.9 (2.0) | -4.9 (2.1)
  Day 8 predose PM | -3.3 (2.9) | -4.1 (2.1) | -3.0 (2.1)
  Day 9 predose AM | 0.6 (2.1) | -4.3 (1.5) | -1.6 (1.5)
  Day 10 predose AM | 0.1 (2.4) | -3.7 (1.7) | -5.0 (1.8)
  Day 11 predose AM | 2.2 (2.5) | -6.4 (1.8) | -3.1 (1.9)
  Day 12 predose AM | -1.1 (2.0) | -3.5 (1.5) | -5.6 (1.5)
  Day 13 predose AM | 0.1 (2.2) | -4.8 (1.6) | -4.4 (1.6)
  Day 13 postdose AM: 1 hour | -2.0 (2.1) | -11.0 (1.6) | -10.5 (1.6)
  Day 13 postdose AM: 4 hour | -2.5 (2.9) | -8.6 (2.1) | -9.0 (2.2)
  Day 13 predose PM | 0.1 (2.7) | -7.8 (2.0) | -7.0 (2.0)
  Day 14 predose AM | -4.4 (3.1) | -6.1 (2.3) | -4.1 (2.3)
  Day 15/Discharge | -0.9 (2.4) | -3.5 (1.8) | -1.6 (1.8)
  Day 21/Follow-Up | 0.1 (1.8) | -0.7 (1.3) | 0.3 (1.3)
  Day 42/End of Trial | 0.7 (3.3) | 2.8 (2.4) | 1.5 (2.4)
Statistical Analysis 1: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, post-dose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.6, 95% CI 2-sided [-8.9 to 3.8], Standard Error of Mean 3.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, post-dose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.0, 95% CI 2-sided [-8.4 to 4.5], Standard Error of Mean 3.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, post-dose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.9, 95% CI 2-sided [-9.2 to 3.4], Standard Error of Mean 3.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, post-dose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -7.1, 95% CI 2-sided [-13.5 to -0.6], Standard Error of Mean 3.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, post-dose AM 8 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.5, 95% CI 2-sided [-11.5 to 0.6], Standard Error of Mean 2.9 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, post-dose AM 8 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.6, 95% CI 2-sided [-10.8 to 1.5], Standard Error of Mean 3.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, pre-dose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.6, 95% CI 2-sided [-9.4 to 2.2], Standard Error of Mean 2.8 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, pre-dose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.1, 95% CI 2-sided [-8.0 to 3.7], Standard Error of Mean 2.8 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, post-dose PM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.0, 95% CI 2-sided [-13.8 to 3.9], Standard Error of Mean 4.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 10: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, post-dose PM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.7, 95% CI 2-sided [-11.7 to 6.2], Standard Error of Mean 4.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 2, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.4, 95% CI 2-sided [-9.7 to 0.9], Standard Error of Mean 2.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 12: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 2, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.1, 95% CI 2-sided [-8.5 to 2.2], Standard Error of Mean 2.6 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 2, post-dose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -6.7, 95% CI 2-sided [-13.1 to -0.3], Standard Error of Mean 3.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 14: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 2, post-dose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.3, 95% CI 2-sided [-11.8 to 1.2], Standard Error of Mean 3.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 2, post-dose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.4, 95% CI 2-sided [-14.2 to 3.5], Standard Error of Mean 4.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 16: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 2, post-dose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -8.5, 95% CI 2-sided [-17.5 to 0.5], Standard Error of Mean 4.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 2, pre-dose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.7, 95% CI 2-sided [-11.6 to 0.2], Standard Error of Mean 2.9 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 18: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 2, pre-dose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.6, 95% CI 2-sided [-10.6 to 1.5], Standard Error of Mean 2.9 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 2, post-dose PM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.5, 95% CI 2-sided [-7.4 to 6.4], Standard Error of Mean 3.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 20: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 2, post-dose PM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.3, 95% CI 2-sided [-9.3 to 4.7], Standard Error of Mean 3.4 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 2, post-dose PM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.4, 95% CI 2-sided [-9.4 to 4.6], Standard Error of Mean 3.4 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 22: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 2, post-dose PM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.5, 95% CI 2-sided [-8.7 to 5.6], Standard Error of Mean 3.4 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 3, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.2, 95% CI 2-sided [-6.2 to 6.7], Standard Error of Mean 3.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 24: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 3, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.3, 95% CI 2-sided [-6.2 to 6.8], Standard Error of Mean 3.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 25: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 3, post-dose PM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.5, 95% CI 2-sided [-6.4 to 9.4], Standard Error of Mean 3.8 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 26: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 3, post-dose PM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.3, 95% CI 2-sided [-9.3 to 6.8], Standard Error of Mean 3.9 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 27: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 4, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.3, 95% CI 2-sided [-10.0 to 1.4], Standard Error of Mean 2.8 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 28: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 4, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.5, 95% CI 2-sided [-10.3 to 1.3], Standard Error of Mean 2.8 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 29: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 5, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.4, 95% CI 2-sided [-8.2 to 3.3], Standard Error of Mean 2.8 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 30: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 5, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -7.1, 95% CI 2-sided [-13.0 to -1.3], Standard Error of Mean 2.8 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 31: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 6, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.8, 95% CI 2-sided [-7.7 to 2.2], Standard Error of Mean 2.4 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 32: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 6, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.7, 95% CI 2-sided [-9.7 to 0.3], Standard Error of Mean 2.4 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 33: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.1, 95% CI 2-sided [-11.6 to 3.5], Standard Error of Mean 3.6 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 34: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.3, 95% CI 2-sided [-12.0 to 3.3], Standard Error of Mean 3.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 35: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, post-dose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.3, 95% CI 2-sided [-10.6 to 1.9], Standard Error of Mean 3.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 36: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, post-dose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.7, 95% CI 2-sided [-12.0 to 0.7], Standard Error of Mean 3.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 37: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, post-dose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.0, 95% CI 2-sided [-8.3 to 10.3], Standard Error of Mean 4.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 38: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, post-dose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.2, 95% CI 2-sided [-9.2 to 9.7], Standard Error of Mean 4.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 39: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 8, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.6, 95% CI 2-sided [-11.5 to 2.3], Standard Error of Mean 3.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 40: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 8, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.9, 95% CI 2-sided [-9.9 to 4.2], Standard Error of Mean 3.4 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 41: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 8, post-dose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -9.3, 95% CI 2-sided [-15.5 to -3.0], Standard Error of Mean 3.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 42: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 8, post-dose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -8.3, 95% CI 2-sided [-14.6 to -1.9], Standard Error of Mean 3.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 43: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 8, post-dose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.3, 95% CI 2-sided [-12.6 to 2.0], Standard Error of Mean 3.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 44: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 8, post-dose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.3, 95% CI 2-sided [-8.7 to 6.1], Standard Error of Mean 3.6 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 45: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 8, pre-dose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.7, 95% CI 2-sided [-8.2 to 6.7], Standard Error of Mean 3.6 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 46: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 8, pre-dose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.3, 95% CI 2-sided [-7.3 to 7.9], Standard Error of Mean 3.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 47: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 9, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.9, 95% CI 2-sided [-10.3 to 0.6], Standard Error of Mean 2.6 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 48: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 9, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.2, 95% CI 2-sided [-7.7 to 3.4], Standard Error of Mean 2.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 49: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 10, pre-dose; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.9, 95% CI 2-sided [-10.0 to 2.3], Standard Error of Mean 3.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 50: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 10, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.1, 95% CI 2-sided [-11.4 to 1.2], Standard Error of Mean 3.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 51: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 11, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -8.7, 95% CI 2-sided [-15.2 to -2.2], Standard Error of Mean 3.2 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 52: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 11, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.3, 95% CI 2-sided [-12.0 to 1.3], Standard Error of Mean 3.2 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 53: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 12, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.4, 95% CI 2-sided [-7.6 to 2.8], Standard Error of Mean 2.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 54: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 12, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.5, 95% CI 2-sided [-9.7 to 0.8], Standard Error of Mean 2.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 55: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 13, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.9, 95% CI 2-sided [-10.7 to 0.8], Standard Error of Mean 2.8 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 56: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 13, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.6, 95% CI 2-sided [-10.4 to 1.3], Standard Error of Mean 2.8 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 57: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 13, post-dose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -9.0, 95% CI 2-sided [-14.6 to -3.4], Standard Error of Mean 2.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 58: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 13, post-dose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -8.5, 95% CI 2-sided [-14.2 to -2.8], Standard Error of Mean 2.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 59: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 13, post-dose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -6.2, 95% CI 2-sided [-13.8 to 1.5], Standard Error of Mean 3.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 60: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 13, post-dose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -6.5, 95% CI 2-sided [-14.3 to 1.2], Standard Error of Mean 3.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 61: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 13, pre-dose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = -8.0, 95% CI 2-sided [-15.0 to -1.0], Standard Error of Mean 3.4 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 62: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 13, pre-dose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = -7.1, 95% CI 2-sided [-14.2 to 0], Standard Error of Mean 3.4 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 63: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.7, 95% CI 2-sided [-9.8 to 6.4], Standard Error of Mean 3.9 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 64: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.3, 95% CI 2-sided [-8.0 to 8.5], Standard Error of Mean 4.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 65: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 15, Discharge; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.6, 95% CI 2-sided [-9.0 to 3.7], Standard Error of Mean 3.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 66: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 15, Discharge; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.7, 95% CI 2-sided [-7.1 to 5.8], Standard Error of Mean 3.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 67: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 21, Follow-up; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.8, 95% CI 2-sided [-5.5 to 3.9], Standard Error of Mean 2.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 68: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 21, Follow-up; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.2, 95% CI 2-sided [-4.6 to 4.9], Standard Error of Mean 2.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 69: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 42, End of trial; Test type: Other — No statistical testing was performed; Least squares mean difference = 2.1, 95% CI 2-sided [-6.5 to 10.7], Standard Error of Mean 4.2 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 70: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 42, End of trial; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.8, 95% CI 2-sided [-7.9 to 9.6], Standard Error of Mean 4.2 — [estimate comment as in outcome 1, analysis 2]

3. Primary Outcome: Change From Study Baseline Over Time in Supine Pulse
Time Frame: as for outcome 1
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment.
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
bpm
  Study Baseline (Day 1 predose AM) | 70.3 (13.7) | 70.3 (10.9) | 70.0 (10.3)
  Day 1 postdose AM: 1 hour | 1.0 (4.1) | 7.2 (3.1) | 10.2 (3.1)
  Day 1 postdose AM: 4 hour | 4.3 (3.4) | 4.3 (2.7) | 8.8 (2.7)
  Day 1 postdose AM: 8 hour | 2.8 (2.8) | 2.6 (2.2) | 4.5 (2.2)
  Day 1 predose PM | 0 (2.7) | 5.1 (2.1) | 5.3 (2.1)
  Day 1 postdose PM: 1 hour | 2.3 (2.8) | 4.6 (2.2) | 3.7 (2.2)
  Day 2 predose AM | -2.6 (2.3) | -1.7 (1.8) | -1.9 (1.8)
  Day 2 postdose AM: 1 hour | 7.0 (4.1) | 9.5 (3.1) | 11.3 (3.1)
  Day 2 postdose AM: 4 hour | 3.2 (3.0) | 6.5 (2.3) | 10.2 (2.3)
  Day 2 predose PM | 7.9 (2.7) | 6.5 (2.1) | 6.6 (2.1)
  Day 2 postdose PM: 1 hour | 7.2 (3.6) | 7.3 (2.8) | 7.0 (2.8)
  Day 2 postdose PM: 4 hour | 1.9 (2.4) | 3.0 (1.8) | 4.8 (1.8)
  Day 3 predose AM | 0.2 (2.3) | -1.2 (1.8) | -0.2 (1.8)
  Day 3 postdose PM: 4 hour | 3.0 (2.9) | 0.7 (2.2) | 5.2 (2.2)
  Day 4 predose AM | -4.1 (2.6) | 2.8 (2.0) | 0.9 (2.0)
  Day 5 predose AM | -3.3 (2.3) | -0.4 (1.8) | -0.6 (1.8)
  Day 6 predose AM | -0.8 (2.9) | 1.5 (2.3) | -1.5 (2.3)
  Day 7 predose AM | -4.0 (2.5) | 1.1 (2.0) | 1.0 (2.0)
  Day 7 postdose AM: 1 hour | 0.2 (4.2) | 9.5 (3.2) | 13.2 (3.2)
  Day 7 postdose AM: 4 hour | -2.6 (2.6) | 4.4 (2.0) | 8.8 (2.0)
  Day 8 predose AM | -2.8 (2.6) | -0.9 (2.0) | 1.3 (2.0)
  Day 8 postdose AM: 1 hour | 2.7 (3.8) | 12.4 (2.9) | 12.3 (2.9)
  Day 8 postdose AM: 4 hour | -0.6 (3.0) | 7.1 (2.3) | 7.7 (2.3)
  Day 8 predose PM | 2.7 (3.2) | 6.0 (2.5) | 5.7 (2.5)
  Day 9 predose AM | -1.8 (2.9) | -0.3 (2.3) | 0.5 (2.3)
  Day 10 predose AM | -3.0 (3.2) | 1.3 (2.4) | 2.1 (2.4)
  Day 11 predose AM | 2.2 (3.6) | 0.7 (2.8) | 1.4 (2.8)
  Day 12 predose AM | -0.6 (4.0) | 2.3 (3.1) | 0.6 (3.1)
  Day 13 predose AM | -0.2 (3.6) | 0.8 (2.8) | -0.1 (2.8)
  Day 13 postdose AM: 1 hour | 0.3 (3.2) | 7.3 (2.5) | 10.2 (2.5)
  Day 13 postdose AM: 4 hour | -0.8 (2.5) | 4.8 (2.0) | 6.4 (2.0)
  Day 13 predose PM | 5.0 (3.0) | 4.5 (2.3) | 7.0 (2.3)
  Day 14 predose AM | -3.1 (3.0) | 0.7 (2.3) | 0.1 (2.3)
  Day 15/Discharge | 1.1 (2.9) | 0.7 (2.3) | 1.5 (2.3)
  Day 21/Follow-Up | -1.3 (4.1) | -2.0 (3.2) | 5.4 (3.2)
  Day 42/End of Trial | 0.4 (3.6) | 0.6 (2.8) | 1.2 (2.8)
Statistical Analysis 1: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, post-dose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 6.2, 95% CI 2-sided [-4.4 to 16.8], Standard Error of Mean 5.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, post-dose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 9.1, 95% CI 2-sided [-1.5 to 19.8], Standard Error of Mean 5.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, post-dose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 0, 95% CI 2-sided [-9.0 to 9.0], Standard Error of Mean 4.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, post-dose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 4.4, 95% CI 2-sided [-4.6 to 13.4], Standard Error of Mean 4.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, post-dose AM 8 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.2, 95% CI 2-sided [-7.5 to 7.1], Standard Error of Mean 3.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, post-dose AM 8 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.6, 95% CI 2-sided [-5.7 to 8.9], Standard Error of Mean 3.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, pre-dose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = 5.1, 95% CI 2-sided [-2.0 to 12.1], Standard Error of Mean 3.4 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, pre-dose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = 5.2, 95% CI 2-sided [-1.8 to 12.3], Standard Error of Mean 3.4 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, post-dose PM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 2.3, 95% CI 2-sided [-5.1 to 9.6], Standard Error of Mean 3.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 10: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, post-dose PM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.3, 95% CI 2-sided [-6.0 to 8.7], Standard Error of Mean 3.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 2, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.0, 95% CI 2-sided [-5.0 to 6.9], Standard Error of Mean 2.9 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 12: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 2, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.7, 95% CI 2-sided [-5.3 to 6.6], Standard Error of Mean 2.9 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 2, post-dose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 2.5, 95% CI 2-sided [-8.1 to 13.2], Standard Error of Mean 5.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 14: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 2, post-dose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 4.3, 95% CI 2-sided [-6.3 to 15.0], Standard Error of Mean 5.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 2, post-dose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 3.3, 95% CI 2-sided [-4.6 to 11.2], Standard Error of Mean 3.8 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 16: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 2, post-dose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 7.0, 95% CI 2-sided [-1.0 to 14.9], Standard Error of Mean 3.8 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 2, pre-dose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.3, 95% CI 2-sided [-8.5 to 5.9], Standard Error of Mean 3.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 18: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 2, pre-dose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.3, 95% CI 2-sided [-8.5 to 5.9], Standard Error of Mean 3.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 2, post-dose PM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.1, 95% CI 2-sided [-9.2 to 9.5], Standard Error of Mean 4.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 20: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 2, post-dose PM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.2, 95% CI 2-sided [-9.5 to 9.2], Standard Error of Mean 4.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 2, post-dose PM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.2, 95% CI 2-sided [-5.1 to 7.4], Standard Error of Mean 3.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 22: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 2, post-dose PM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 2.9, 95% CI 2-sided [-3.4 to 9.2], Standard Error of Mean 3.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 3, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.4, 95% CI 2-sided [-7.5 to 4.8], Standard Error of Mean 3.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 24: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 3, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.4, 95% CI 2-sided [-6.5 to 5.8], Standard Error of Mean 3.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 25: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 3, post-dose PM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.3, 95% CI 2-sided [-9.9 to 5.3], Standard Error of Mean 3.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 26: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 3, post-dose PM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 2.2, 95% CI 2-sided [-5.4 to 9.8], Standard Error of Mean 3.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 27: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 4, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 7.0, 95% CI 2-sided [0.2 to 13.7], Standard Error of Mean 3.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 28: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 4, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 5.0, 95% CI 2-sided [-1.7 to 11.8], Standard Error of Mean 3.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 29: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 5, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 2.9, 95% CI 2-sided [-3.1 to 9.0], Standard Error of Mean 2.9 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 30: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 5, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 2.6, 95% CI 2-sided [-3.4 to 8.7], Standard Error of Mean 2.9 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 31: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 6, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 2.3, 95% CI 2-sided [-5.4 to 10.0], Standard Error of Mean 3.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 32: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 6, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.7, 95% CI 2-sided [-8.4 to 7.0], Standard Error of Mean 3.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 33: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 5.1, 95% CI 2-sided [-1.6 to 11.8], Standard Error of Mean 3.2 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 34: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 5.0, 95% CI 2-sided [-1.7 to 11.7], Standard Error of Mean 3.2 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 35: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, post-dose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 9.3, 95% CI 2-sided [-1.6 to 20.2], Standard Error of Mean 5.2 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 36: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, post-dose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 13.0, 95% CI 2-sided [2.1 to 23.9], Standard Error of Mean 5.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 37: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, post-dose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 7.1, 95% CI 2-sided [0.2 to 13.9], Standard Error of Mean 3.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 38: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, post-dose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 11.5, 95% CI 2-sided [4.6 to 18.3], Standard Error of Mean 3.3 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 39: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 8, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.9, 95% CI 2-sided [-4.8 to 8.6], Standard Error of Mean 3.2 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 40: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 8, pre-dose; Test type: Other — No statistical testing was performed; Least squares mean difference = 4.1, 95% CI 2-sided [-2.6 to 10.8], Standard Error of Mean 3.2 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 41: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 8, post-dose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 9.7, 95% CI 2-sided [-0.1 to 19.6], Standard Error of Mean 4.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 42: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 8, post-dose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 9.6, 95% CI 2-sided [-0.3 to 19.4], Standard Error of Mean 4.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 43: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 8, post-dose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 7.8, 95% CI 2-sided [0 to 15.5], Standard Error of Mean 3.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 44: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 8, post-dose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 8.3, 95% CI 2-sided [0.6 to 16.1], Standard Error of Mean 3.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 45: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 8, pre-dose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = 3.3, 95% CI 2-sided [-5.1 to 11.7], Standard Error of Mean 4.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 46: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 8, pre-dose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = 3.0, 95% CI 2-sided [-5.4 to 11.3], Standard Error of Mean 4.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 47: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 9, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.5, 95% CI 2-sided [-6.1 to 9.1], Standard Error of Mean 3.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 48: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 9, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 2.3, 95% CI 2-sided [-5.3 to 9.9], Standard Error of Mean 3.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 49: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 10, pre-dose; Test type: Other — No statistical testing was performed; Least squares mean difference = 4.3, 95% CI 2-sided [-4.0 to 12.6], Standard Error of Mean 4.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 50: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 10, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 5.1, 95% CI 2-sided [-3.2 to 13.4], Standard Error of Mean 4.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 51: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 11, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.5, 95% CI 2-sided [-11.0 to 8.0], Standard Error of Mean 4.6 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 52: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 11, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.9, 95% CI 2-sided [-10.3 to 8.6], Standard Error of Mean 4.6 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 53: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 12, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 2.9, 95% CI 2-sided [-7.7 to 13.4], Standard Error of Mean 5.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 54: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 12, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.2, 95% CI 2-sided [-9.4 to 11.8], Standard Error of Mean 5.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 55: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 13, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.0, 95% CI 2-sided [-8.4 to 10.3], Standard Error of Mean 4.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 56: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 13, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.1, 95% CI 2-sided [-9.3 to 9.4], Standard Error of Mean 4.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 57: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 13, post-dose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 7.0, 95% CI 2-sided [-1.3 to 15.3], Standard Error of Mean 4.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 58: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 13, post-dose AM 1 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 9.9, 95% CI 2-sided [1.6 to 18.2], Standard Error of Mean 4.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 59: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 13, post-dose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 5.6, 95% CI 2-sided [-1.0 to 12.3], Standard Error of Mean 3.2 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 60: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 13, post-dose AM 4 hour; Test type: Other — No statistical testing was performed; Least squares mean difference = 7.2, 95% CI 2-sided [0.5 to 13.9], Standard Error of Mean 3.2 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 61: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 13, pre-dose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.5, 95% CI 2-sided [-8.4 to 7.4], Standard Error of Mean 3.8 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 62: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 13, pre-dose PM; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.9, 95% CI 2-sided [-6.0 to 9.9], Standard Error of Mean 3.8 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 63: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 3.9, 95% CI 2-sided [-4.0 to 11.8], Standard Error of Mean 3.8 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 64: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, pre-dose AM; Test type: Other — No statistical testing was performed; Least squares mean difference = 3.3, 95% CI 2-sided [-4.6 to 11.2], Standard Error of Mean 3.8 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 65: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 15, Discharge; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.3, 95% CI 2-sided [-8.0 to 7.3], Standard Error of Mean 3.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 66: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 15, Discharge; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.5, 95% CI 2-sided [-7.2 to 8.1], Standard Error of Mean 3.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 67: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 21, Follow-up; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.7, 95% CI 2-sided [-11.5 to 10.2], Standard Error of Mean 5.2 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 68: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 21, Follow-up; Test type: Other — No statistical testing was performed; Least squares mean difference = 6.7, 95% CI 2-sided [-4.1 to 17.5], Standard Error of Mean 5.2 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 69: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 42, End of trial; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.3, 95% CI 2-sided [-9.1 to 9.6], Standard Error of Mean 4.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 70: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 42, End of trial; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.8, 95% CI 2-sided [-8.5 to 10.2], Standard Error of Mean 4.5 — [estimate comment as in outcome 1, analysis 2]

4. Primary Outcome: Percentage of Participants With Postdose Supine Blood Pressure Less Than 130/80 mmHg Over Time
Time Frame: Baseline, Days 1-14, Day 15, 21, 42
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
percentage of participants
  Baseline | 33.3 | 80.0 | 60.0
  Day 1 | 100 | 100 | 100
  Day 2 | 66.7 | 100 | 100
  Day 3 | 66.7 | 100 | 90.0
  Day 4 | 50.0 | 100 | 90.0
  Day 5 | 50.0 | 70.0 | 90.0
  Day 6 | 66.7 | 90.0 | 90.0
  Day 7 | 50.0 | 90.0 | 90.0
  Day 8 | 83.3 | 90.0 | 100
  Day 9 | 33.3 | 100 | 70.0
  Day 10 | 33.3 | 100 | 70.0
  Day 11 | 50.0 | 100 | 70.0
  Day 12 | 50.0 | 90.0 | 80.0
  Day 13 | 66.7 | 100 | 100
  Day 14 | 50.0 | 90.0 | 80.0
  Day 15 / Discharge | 33.3 | 100 | 70.0
  Day 21 / Follow-Up | 50.0 | 80.0 | 50.0
  Day 42 / End of Trial | 33.3 | 40.0 | 60.0

5. Primary Outcome: Orthostatic Systolic Blood Pressure Over Time
Description: An orthostatic measurement is obtained by subtracting the supine measurement from the standing measurement.
Time Frame: Days -1, 1, 2, 7, 8, 13: 1 and 4 hour AM; Days -1, 1, 2, 8, 13: 0 hour PM; Days -1, 1, 2: 1 hour PM; Days 1, 2, 7, 8, 13: 0 hour AM; Day 1: 8 hour AM; Days 1, 2: 4 hour PM
Population: Safety Population: participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
mmHg
  Day -1, 1 hour AM | -0.8 (11.9) | 2.0 (12.1) | 5.6 (11.5)
  Day -1, 4 hour AM | 0.3 (6.4) | 2.9 (9.9) | 2.3 (11.5)
  Day -1, 0 hour PM | 3.0 (10.5) | 1.7 (12.4) | -0.1 (7.3)
  Day -1, 1 hour PM | 3.8 (9.0) | 5.3 (13.8) | 3.1 (11.5)
  Day 1, 0 hour AM | 1.3 (9.6) | 5.2 (11.8) | 3.7 (12.7)
  Day 1, 1 hour AM | 9.7 (7.9) | 3.7 (15.8) | 2.5 (11.5)
  Day 1, 4 hour AM | 3.0 (14.6) | 12.1 (11.3) | 5.8 (8.3)
  Day 1, 8 hour AM | 5.3 (6.4) | 4.7 (12.4) | 5.1 (11.5)
  Day 1, 0 hour PM | 10.2 (10.5) | 4.1 (17.0) | 0.2 (10.3)
  Day 1, 1 hour PM | 5.7 (10.2) | 0.7 (18.0) | 4.1 (11.4)
  Day 1, 4 hour PM | 4.3 (14.4) | 0.4 (14.8) | 6.4 (5.3)
  Day 2, 0 hour AM | -2.7 (11.0) | 2.5 (13.5) | 1.1 (10.3)
  Day 2, 1 hour AM | -4.7 (15.0) | 2.9 (8.5) | 2.2 (8.6)
  Day 2, 4 hour AM | -1.7 (11.4) | 5.8 (6.8) | 4.6 (10.6)
  Day 2, 0 Hour PM | -6.0 (14.9) | 6.6 (11.9) | 2.3 (10.4)
  Day 2, 1 hour PM | 2.7 (14.4) | 5.0 (14.3) | 0.5 (14.0)
  Day 2, 4 hour PM | 0.8 (6.8) | -0.7 (18.9) | 7.1 (13.1)
  Day 7, 0 hour AM | 1.0 (7.6) | 2.5 (19.1) | 4.9 (10.7)
  Day 7, 1 hour AM | -2.0 (6.8) | 6.3 (11.7) | -2.5 (8.0)
  Day 7, 4 hour AM | -1.2 (10.8) | 4.7 (11.3) | 4.7 (14.1)
  Day 8, 0 hour AM | -4.0 (13.7) | 6.5 (11.9) | -1.1 (5.7)
  Day 8, 1 hour AM | -2.5 (8.5) | 5.9 (14.7) | 1.7 (12.6)
  Day 8, 4 hour AM | 1.0 (12.3) | 2.9 (10.3) | -1.7 (16.0)
  Day 8, 0 hour PM | 1.0 (8.4) | 5.0 (9.7) | 4.2 (8.8)
  Day 13, 0 hour AM | -2.0 (5.2) | 6.2 (13.7) | 1.3 (7.4)
  Day 13, 1 hour AM | -1.5 (12.8) | 8.3 (13.7) | 1.4 (12.1)
  Day 13, 4 hour AM | 0.8 (7.4) | 4.1 (10.9) | 2.2 (11.7)
  Day 13, 0 hour PM | 3.8 (9.1) | 4.8 (14.2) | 3.2 (10.3)

6. Primary Outcome: Orthostatic Diastolic Blood Pressure Over Time
Description: An orthostatic measurement is obtained by subtracting the supine measurement from the standing measurement.
Time Frame: as for outcome 5
Population: Safety Population: participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
mmHg
  Day -1, 1 hour AM | 1.8 (3.0) | 3.3 (6.8) | 6.3 (5.9)
  Day -1, 4 hour AM | -0.5 (5.1) | 3.6 (8.2) | 5.5 (6.4)
  Day -1, 0 hour PM | 8.2 (4.6) | 4.2 (5.6) | 3.4 (4.4)
  Day -1, 1 hour PM | 5.7 (4.6) | 4.0 (6.8) | 4.5 (4.3)
  Day 1, 0 hour AM | 3.3 (5.2) | 4.2 (4.4) | 5.4 (4.6)
  Day 1, 1 hour AM | 5.3 (8.9) | 2.9 (5.1) | 3.4 (5.9)
  Day 1, 4 hour AM | 4.2 (4.1) | 6.1 (5.8) | 7.0 (5.0)
  Day 1, 8 hour AM | 5.3 (1.9) | 3.6 (4.5) | 4.9 (6.0)
  Day 1, 0 hour PM | 10.0 (6.8) | 2.8 (6.3) | 5.1 (6.2)
  Day 1, 1 hour PM | 3.0 (4.3) | 5.2 (9.2) | 5.1 (4.3)
  Day 1, 4 hour PM | 6.8 (4.2) | 3.4 (7.3) | 7.7 (4.9)
  Day 2, 0 hour AM | 2.7 (2.0) | 3.3 (5.2) | 3.3 (6.0)
  Day 2, 1 hour AM | 3.0 (4.1) | 1.8 (5.8) | 5.2 (3.2)
  Day 2, 4 hour AM | 0.5 (2.4) | 3.8 (3.5) | 5.7 (5.3)
  Day 2, 0 Hour PM | -2.7 (10.2) | 3.2 (7.4) | 4.7 (5.2)
  Day 2, 1 hour PM | 2.3 (5.6) | 0.9 (6.1) | 5.3 (5.1)
  Day 2, 4 hour PM | 5.8 (4.3) | 1.3 (10.0) | 8.7 (7.5)
  Day 7, 0 hour AM | 2.3 (3.4) | 2.9 (7.9) | 5.6 (6.2)
  Day 7, 1 hour AM | 1.8 (2.9) | 3.7 (5.5) | 2.4 (3.5)
  Day 7, 4 hour AM | 7.3 (9.0) | 4.8 (7.4) | 3.2 (6.5)
  Day 8, 0 hour AM | 3.3 (6.1) | 6.2 (7.1) | 4.8 (5.5)
  Day 8, 1 hour AM | -1.3 (8.9) | 2.2 (8.4) | 3.8 (6.7)
  Day 8, 4 hour AM | 4.0 (2.6) | 1.9 (7.3) | 1.2 (7.3)
  Day 8, 0 hour PM | 5.0 (2.6) | 3.8 (4.5) | 4.2 (4.0)
  Day 13, 0 hour AM | 2.7 (5.1) | 4.0 (6.8) | 3.9 (4.1)
  Day 13, 1 hour AM | 3.3 (4.3) | 5.8 (4.7) | 5.0 (7.1)
  Day 13, 4 hour AM | 0.7 (4.5) | 3.7 (4.3) | 5.4 (7.7)
  Day 13, 0 hour PM | 4.0 (3.2) | 5.1 (6.3) | 3.9 (3.8)

7. Primary Outcome: Orthostatic Pulse Over Time
Description: An orthostatic measurement is obtained by subtracting the supine measurement from the standing measurement.
Time Frame: as for outcome 5
Population: Safety Population: participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
bpm
  Day -1, 1 hour AM | 9.2 (6.4) | 9.2 (4.3) | 10.2 (8.8)
  Day -1, 4 hour AM | 4.7 (9.8) | 10.9 (5.8) | 9.5 (8.3)
  Day -1, 0 hour PM | 15.3 (15.0) | 10.1 (4.7) | 9.8 (4.9)
  Day -1, 1 hour PM | 11.3 (3.9) | 11.0 (4.3) | 11.4 (6.0)
  Day 1, 0 hour AM | 4.8 (10.4) | 8.8 (4.3) | 10.3 (7.7)
  Day 1, 1 hour AM | 8.7 (6.6) | 9.7 (5.9) | 12.9 (6.9)
  Day 1, 4 hour AM | 7.7 (7.4) | 11.0 (6.1) | 10.1 (8.4)
  Day 1, 8 hour AM | 10.0 (4.7) | 9.9 (6.3) | 10.5 (4.6)
  Day 1, 0 hour PM | 14.8 (9.9) | 9.1 (6.6) | 7.7 (4.1)
  Day 1, 1 hour PM | 9.3 (6.2) | 10.8 (7.2) | 11.1 (6.6)
  Day 1, 4 hour PM | 16.5 (12.7) | 14.5 (7.2) | 16.5 (10.0)
  Day 2, 0 hour AM | 9.0 (3.0) | 10.4 (7.0) | 10.5 (4.7)
  Day 2, 1 hour AM | 6.5 (6.0) | 11.2 (8.7) | 10.7 (5.8)
  Day 2, 4 hour AM | 11.2 (9.2) | 8.4 (6.5) | 8.8 (6.2)
  Day 2, 0 Hour PM | 6.0 (8.6) | 8.6 (5.8) | 9.0 (4.2)
  Day 2, 1 hour PM | 10.0 (5.4) | 9.4 (6.8) | 7.9 (4.6)
  Day 2, 4 hour PM | 10.8 (6.3) | 15.9 (8.6) | 13.6 (7.1)
  Day 7, 0 hour AM | 10.8 (5.2) | 7.1 (8.5) | 9.7 (4.6)
  Day 7, 1 hour AM | 11.5 (6.3) | 9.5 (6.6) | 10.1 (7.9)
  Day 7, 4 hour AM | 10.8 (3.3) | 8.7 (2.6) | 9.6 (4.7)
  Day 8, 0 hour AM | 10.3 (8.3) | 8.6 (8.6) | 9.5 (7.8)
  Day 8, 1 hour AM | 5.3 (9.3) | 9.5 (8.7) | 10.5 (3.3)
  Day 8, 4 hour AM | 10.7 (7.4) | 8.1 (7.8) | 7.3 (6.1)
  Day 8, 0 hour PM | 9.3 (3.6) | 9.6 (5.6) | 8.9 (4.7)
  Day 13, 0 hour AM | 7.8 (14.9) | 9.1 (8.6) | 10.9 (5.9)
  Day 13, 1 hour AM | 11.0 (4.6) | 7.9 (6.0) | 11.2 (7.5)
  Day 13, 4 hour AM | 14.5 (8.1) | 9.1 (6.0) | 11.5 (5.9)
  Day 13, 0 hour PM | 9.3 (3.4) | 9.3 (4.6) | 11.2 (4.3)

8. Primary Outcome: Change From Time-Matched Baseline Over Time in Ambulatory Blood Pressure Monitoring (ABPM) 24-hour Averages of Systolic Blood Pressure
Description: 24-hour average is the average of ABPM assessments over 24 hour intervals from the time of dosing. Time-matched baseline is the 24 hours average during Day -1.
Time Frame: Time Matched Baseline (Day -1), Days 1, 7, and 14
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Groups:
- IW-1973 40 mg Total Daily Dose (Overall): IW-1973 40 mg BID/QD:
  IW-973 20 mg oral tablet taken in AM and 20 mg oral tablet taken in PM on Days 1-7. IW-1973 40 mg oral tablet taken QD in AM and placebo oral tablet taken QD in PM on Days 8-14.
  IW-1973 40 mg QD/QD:
  IW-1973 40 mg oral tablet taken QD in AM and placebo taken QD in PM on Days 1-14.
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD | IW-1973 40 mg Total Daily Dose (Overall)
Number analyzed (Participants) | 6 | 10 | 10 | 20
mmHg
  Time Matched Baseline (Day -1) | 132.34 (8.22) | 126.40 (11.07) | 129.00 (6.48) | 127.70 (8.93)
  Change at Day 1 | -0.60 (2.39) | -3.92 (1.84) | -3.15 (1.81) | -3.53 (1.29)
  Change at Day 7 | -3.54 (2.68) | -6.77 (2.07) | -3.03 (2.04) | -4.90 (1.45)
  Change at Day 14 | -4.87 (3.17) | -7.58 (2.59) | -6.74 (2.39) | -7.16 (1.75)
Statistical Analysis 1: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.32, 95% CI 2-sided [-9.68 to 3.04], Standard Error of Mean 3.07 — Least Squares mean difference and associated 95% CI is from an ANCOVA model with treatment as fixed effect and baseline as covariate. Standard Error of the Mean=Standard Error of the LS Mean Difference
Statistical Analysis 2: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.55, 95% CI 2-sided [-8.76 to 3.66], Standard Error of Mean 2.99 — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs IW-1973 40 mg Total Daily Dose (Overall); Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.93, 95% CI 2-sided [-8.62 to 2.75], Standard Error of Mean 2.74 — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.23, 95% CI 2-sided [-10.37 to 3.92], Standard Error of Mean 3.44 — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.52, 95% CI 2-sided [-6.46 to 7.49], Standard Error of Mean 3.36 — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs IW-1973 40 mg Total Daily Dose (Overall); Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.36, 95% CI 2-sided [-7.74 to 5.03], Standard Error of Mean 3.08 — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.71, 95% CI 2-sided [-11.46 to 6.04], Standard Error of Mean 4.21 — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.87, 95% CI 2-sided [-10.09 to 6.35], Standard Error of Mean 3.95 — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs IW-1973 40 mg Total Daily Dose (Overall); Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.29, 95% CI 2-sided [-9.93 to 5.35], Standard Error of Mean 3.67 — [estimate comment as in outcome 8, analysis 1]

9. Primary Outcome: Change From Time-Matched Baseline Over Time in ABPM Daytime (12-Hour) Averages of Systolic Blood Pressure
Description: Daytime 12-hour average is the average of ABPM assessments over daytime 12-hour intervals from the time of dosing. Time-matched baseline is the daytime 12 hours average during Day -1.
Time Frame: Time Matched Baseline (Day -1), Days 1, 7, and 14
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
mmHg
  Time Matched Baseline (Day -1) | 136.99 (8.42) | 130.64 (10.82) | 132.28 (7.07)
  Change at Day 1 | -0.74 (2.81) | -7.80 (2.14) | -4.93 (2.12)
  Change at Day 7 | -5.27 (2.89) | -9.09 (2.20) | -3.85 (2.17)
  Change at Day 14 | -6.37 (3.62) | -12.81 (2.92) | -7.40 (2.71)
Statistical Analysis 1: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = -7.06, 95% CI 2-sided [-14.52 to 0.40], Standard Error of Mean 3.60 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.19, 95% CI 2-sided [-11.52 to 3.14], Standard Error of Mean 3.54 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.82, 95% CI 2-sided [-11.47 to 3.83], Standard Error of Mean 3.69 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.42, 95% CI 2-sided [-6.10 to 8.94], Standard Error of Mean 3.63 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = -6.44, 95% CI 2-sided [-16.36 to 3.47], Standard Error of Mean 4.77 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.03, 95% CI 2-sided [-10.44 to 8.38], Standard Error of Mean 4.52 — [estimate comment as in outcome 1, analysis 2]

10. Primary Outcome: Change From Time-Matched Baseline Over Time in ABPM Nighttime (12-Hour) Averages of Systolic Blood Pressure
Description: Nighttime 12-hour average is the average of ABPM assessments over nighttime 12-hour intervals from the time of dosing. Time-matched baseline is the nighttime 12 hours average during Day -1.
Time Frame: Time Matched Baseline (Day -1), Days 1, 7, and 14
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
mmHg
  Time Matched Baseline (Day -1) | 126.76 (9.36) | 121.77 (12.26) | 125.26 (7.24)
  Change at Day 1 | 0.11 (2.55) | -0.11 (1.98) | -1.50 (1.96)
  Change at Day 7 | -1.42 (2.93) | -4.54 (2.28) | -2.25 (2.25)
  Change at Day 14 | -3.25 (3.17) | -2.38 (2.63) | -6.23 (2.44)
Statistical Analysis 1: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.22, 95% CI 2-sided [-6.97 to 6.54], Standard Error of Mean 3.26 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.60, 95% CI 2-sided [-8.24 to 5.03], Standard Error of Mean 3.20 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.12, 95% CI 2-sided [-10.88 to 4.65], Standard Error of Mean 3.74 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.82, 95% CI 2-sided [-8.45 to 6.80], Standard Error of Mean 3.68 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.87, 95% CI 2-sided [-7.84 to 9.58], Standard Error of Mean 4.19 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.98, 95% CI 2-sided [-11.23 to 5.26], Standard Error of Mean 3.96 — [estimate comment as in outcome 1, analysis 2]

11. Primary Outcome: Change From Time-Matched Baseline Over Time in ABPM 4-hour Averages of Systolic Blood Pressure
Description: Postdose is the average of assessments over 4-hour intervals from the time of dosing that day. Time-matched baseline is the corresponding 4-hour average on Day -1.
Time Frame: Time-matched baseline (Day -1), Days 1, 7, 14: 0-4, 4-8, 8-12, 12-16, 16-20, 20-24 hours postdose
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
mmHg
  Time-matched baseline (Day -1): 0-4 hours | 134.45 (8.01) | 128.18 (9.90) | 128.38 (7.33)
  Time-matched baseline (Day -1): 4-8 hours | 136.10 (9.69) | 130.04 (13.15) | 132.53 (6.83)
  Time-matched baseline (Day -1): 8-12 hours | 140.46 (9.12) | 133.67 (11.90) | 135.93 (8.51)
  Time-matched baseline (Day -1): 12-16 hours | 130.31 (9.75) | 124.00 (11.93) | 128.44 (11.32)
  Time-matched baseline (Day -1): 16-20 hours | 120.34 (8.79) | 119.75 (14.51) | 120.41 (11.00)
  Time-matched baseline (Day -1): 20-24 hours | 132.10 (11.62) | 122.77 (9.60) | 128.13 (7.19)
  Day 1, 0-4 hours | -1.61 (3.02) | -7.15 (2.27) | -4.08 (2.27)
  Day 1, 4-8 hours | -0.62 (3.51) | -8.67 (2.70) | -8.89 (2.67)
  Day 1, 8-12 hours | 1.21 (3.80) | -8.14 (2.91) | -1.84 (2.88)
  Day 1, 12-16 hours | -4.83 (3.04) | -1.46 (2.37) | -2.00 (2.34)
  Day 1, 16-20 hours | 3.77 (4.12) | -0.66 (3.19) | -1.08 (3.19)
  Day 1, 20-24 hours | 2.08 (3.04) | 1.27 (2.37) | -0.55 (2.27)
  Day 7, 0-4 hours | -5.14 (3.14) | -10.68 (2.35) | -5.15 (2.35)
  Day 7, 4-8 hours | -6.24 (3.44) | -9.13 (2.65) | -4.07 (2.62)
  Day 7, 8-12 hours | -3.70 (3.65) | -7.93 (2.80) | -2.33 (2.76)
  Day 7, 12-16 hours | -4.46 (3.66) | -5.03 (2.86) | -1.97 (2.82)
  Day 7, 16-20 hours | 2.75 (3.98) | -5.14 (3.08) | -3.74 (3.08)
  Day 7, 20-24 hours | -1.10 (3.74) | -4.94 (2.91) | -0.33 (2.80)
  Day 14, 0-4 hours | -6.67 (3.92) | -13.80 (3.10) | -5.01 (2.90)
  Day 14, 4-8 hours | -7.36 (3.62) | -13.67 (2.95) | -8.53 (2.75)
  Day 14, 8-12 hours | -4.42 (4.41) | -11.43 (3.58) | -8.53 (3.31)
  Day 14, 12-16 hours | -5.28 (4.14) | -3.52 (3.43) | -8.75 (3.18)
  Day 14, 16-20 hours | -1.06 (3.53) | -2.79 (2.89) | -6.61 (2.74)
  Day 14, 20-24 hours | -2.98 (3.82) | -1.00 (3.17) | -1.91 (2.84)
Statistical Analysis 1: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.55, 95% CI 2-sided [-13.51 to 2.41], Standard Error of Mean 3.84 — Least squares mean difference and associated 95% CI are from an ANCOVA model with treatment as fixed effect and baseline as covariate
Statistical Analysis 2: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.47, 95% CI 2-sided [-10.41 to 5.47], Standard Error of Mean 3.83 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -8.05, 95% CI 2-sided [-17.36 to 1.25], Standard Error of Mean 4.49 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -8.28, 95% CI 2-sided [-17.42 to 0.87], Standard Error of Mean 4.41 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -9.34, 95% CI 2-sided [-19.43 to 0.74], Standard Error of Mean 4.86 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.05, 95% CI 2-sided [-12.95 to 6.84], Standard Error of Mean 4.77 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 3.36, 95% CI 2-sided [-4.74 to 11.47], Standard Error of Mean 3.91 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 2.82, 95% CI 2-sided [-5.10 to 10.75], Standard Error of Mean 3.82 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.43, 95% CI 2-sided [-15.23 to 6.37], Standard Error of Mean 5.21 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 10: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.85, 95% CI 2-sided [-15.65 to 5.94], Standard Error of Mean 5.21 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 11: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.81, 95% CI 2-sided [-9.10 to 7.47], Standard Error of Mean 4.00 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 12: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.63, 95% CI 2-sided [-10.42 to 5.16], Standard Error of Mean 3.76 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 13: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.54, 95% CI 2-sided [-13.80 to 2.72], Standard Error of Mean 3.98 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 14: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.01, 95% CI 2-sided [-8.25 to 8.23], Standard Error of Mean 3.97 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 15: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.89, 95% CI 2-sided [-12.01 to 6.23], Standard Error of Mean 4.40 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 16: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 2.17, 95% CI 2-sided [-6.78 to 11.13], Standard Error of Mean 4.32 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 17: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.23, 95% CI 2-sided [-13.93 to 5.47], Standard Error of Mean 4.68 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 18: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.37, 95% CI 2-sided [-8.14 to 10.88], Standard Error of Mean 4.59 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 19: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.57, 95% CI 2-sided [-10.32 to 9.18], Standard Error of Mean 4.70 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 20: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 2.49, 95% CI 2-sided [-7.04 to 12.02], Standard Error of Mean 4.60 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 21: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -7.89, 95% CI 2-sided [-18.33 to 2.55], Standard Error of Mean 5.03 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 22: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -6.49, 95% CI 2-sided [-16.92 to 3.95], Standard Error of Mean 5.03 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 23: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.84, 95% CI 2-sided [-14.03 to 6.35], Standard Error of Mean 4.91 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 24: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.78, 95% CI 2-sided [-8.80 to 10.35], Standard Error of Mean 4.62 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 25: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -7.13, 95% CI 2-sided [-17.79 to 3.53], Standard Error of Mean 5.12 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 26: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.66, 95% CI 2-sided [-8.59 to 11.91], Standard Error of Mean 4.93 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 27: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -6.31, 95% CI 2-sided [-16.17 to 3.55], Standard Error of Mean 4.74 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 28: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.17, 95% CI 2-sided [-10.60 to 8.27], Standard Error of Mean 4.54 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 29: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -7.01, 95% CI 2-sided [-19.13 to 5.11], Standard Error of Mean 5.83 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 30: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.11, 95% CI 2-sided [-15.55 to 7.34], Standard Error of Mean 5.50 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 31: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.77, 95% CI 2-sided [-9.63 to 13.17], Standard Error of Mean 5.48 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 32: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.47, 95% CI 2-sided [-14.25 to 7.31], Standard Error of Mean 5.18 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 33: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.73, 95% CI 2-sided [-11.24 to 7.77], Standard Error of Mean 4.57 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 34: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.55, 95% CI 2-sided [-14.83 to 3.73], Standard Error of Mean 4.46 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 35: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.98, 95% CI 2-sided [-8.85 to 12.81], Standard Error of Mean 5.21 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 36: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.07, 95% CI 2-sided [-8.68 to 10.82], Standard Error of Mean 4.69 — [estimate comment as in outcome 11, analysis 1]

12. Primary Outcome: Change From Time-Matched Baseline Over Time in ABPM 24-hour Averages of Mean Arterial Pressure
Description: as for outcome 8
Time Frame: Time Matched Baseline (Day -1), Days 1, 7, and 14
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD | IW-1973 40 mg Total Daily Dose (Overall)
Number analyzed (Participants) | 6 | 10 | 10 | 20
mmHg
  Time Matched Baseline (Day -1) | 96.44 (8.38) | 90.27 (6.89) | 91.14 (5.54) | 90.71 (6.10)
  Change at Day 1 | -0.68 (1.61) | -2.80 (1.20) | -3.07 (1.19) | -2.94 (0.85)
  Change at Day 7 | -1.84 (1.83) | -5.24 (1.37) | -3.46 (1.35) | -4.35 (0.97)
  Change at Day 14: number analyzed (Participants) | 6 | 9 | 10 | 19
  Change at Day 14 | -1.55 (2.28) | -6.50 (1.79) | -6.05 (1.65) | -6.28 (1.23)
Statistical Analysis 1: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.12, 95% CI 2-sided [-6.38 to 2.15], Standard Error of Mean 2.06 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.39, 95% CI 2-sided [-6.59 to 1.80], Standard Error of Mean 2.02 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs IW-1973 40 mg Total Daily Dose (Overall); Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.26, 95% CI 2-sided [-6.11 to 1.60], Standard Error of Mean 1.86 — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.39, 95% CI 2-sided [-8.25 to 1.47], Standard Error of Mean 2.34 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.61, 95% CI 2-sided [-6.40 to 3.18], Standard Error of Mean 2.31 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs IW-1973 40 mg Total Daily Dose (Overall); Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.50, 95% CI 2-sided [-6.90 to 1.90], Standard Error of Mean 2.12 — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.96, 95% CI 2-sided [-11.22 to 1.31], Standard Error of Mean 3.01 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.50, 95% CI 2-sided [-10.41 to 1.40], Standard Error of Mean 2.84 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs IW-1973 40 mg Total Daily Dose (Overall); Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.73, 95% CI 2-sided [-10.27 to 0.81], Standard Error of Mean 2.67 — [estimate comment as in outcome 8, analysis 1]

13. Primary Outcome: Change From Time-Matched Baseline Over Time in ABPM Daytime (12-hour) Averages of Mean Arterial Pressure
Description: as for outcome 9
Time Frame: Time Matched Baseline (Day -1), Days 1, 7, and 14
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
mmHg
  Time Matched Baseline (Day -1) | 100.09 (7.14) | 93.31 (7.36) | 94.00 (5.54)
  Change at Day 1 | -0.20 (2.24) | -5.07 (1.65) | -5.22 (1.63)
  Change at Day 7 | -2.60 (2.01) | -6.82 (1.48) | -4.75 (1.46)
  Change at Day 14: number analyzed (Participants) | 6 | 9 | 10
  Change at Day 14 | -1.97 (2.50) | -10.71 (1.94) | -7.31 (1.79)
Statistical Analysis 1: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.87, 95% CI 2-sided [-10.80 to 1.06], Standard Error of Mean 2.86 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.02, 95% CI 2-sided [-10.87 to 0.83], Standard Error of Mean 2.82 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.23, 95% CI 2-sided [-9.55 to 1.10], Standard Error of Mean 2.57 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.15, 95% CI 2-sided [-7.40 to 3.11], Standard Error of Mean 2.53 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = -8.74, 95% CI 2-sided [-15.64 to -1.85], Standard Error of Mean 3.31 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.34, 95% CI 2-sided [-11.84 to 1.15], Standard Error of Mean 3.12 — [estimate comment as in outcome 1, analysis 2]

14. Primary Outcome: Change From Time-Matched Baseline Over Time in ABPM Nighttime (12-Hour) Averages of Mean Arterial Pressure
Description: as for outcome 10
Time Frame: Time Matched Baseline (Day -1), Days 1, 7, and 14
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
mmHg
  Time Matched Baseline (Day -1) | 91.93 (10.03) | 86.85 (7.57) | 87.77 (6.37)
  Change at Day 1 | -0.39 (1.67) | -0.84 (1.27) | -1.10 (1.26)
  Change at Day 7 | -0.47 (2.07) | -3.79 (1.57) | -2.20 (1.56)
  Change at Day 14: number analyzed (Participants) | 6 | 9 | 10
  Change at Day 14 | -0.54 (2.46) | -2.42 (1.97) | -4.83 (1.84)
Statistical Analysis 1: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.45, 95% CI 2-sided [-4.86 to 3.96], Standard Error of Mean 2.13 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.71, 95% CI 2-sided [-5.07 to 3.65], Standard Error of Mean 2.10 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.32, 95% CI 2-sided [-8.79 to 2.14], Standard Error of Mean 2.64 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.74, 95% CI 2-sided [-7.14 to 3.67], Standard Error of Mean 2.61 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.88, 95% CI 2-sided [-8.58 to 4.83], Standard Error of Mean 3.22 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.30, 95% CI 2-sided [-10.69 to 2.10], Standard Error of Mean 3.08 — [estimate comment as in outcome 1, analysis 2]

15. Primary Outcome: Change From Time-Matched Baseline Over Time in ABPM 4-hour Averages of Mean Arterial Pressure
Description: as for outcome 11
Time Frame: Time-matched baseline (Day -1), Days 1, 7, 14: 0-4, 4-8, 8-12, 12-16, 16-20, 20-24 hours postdose
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
mmHg
  Time-matched baseline (Day -1): 0-4 hours | 98.10 (5.10) | 91.52 (7.00) | 91.16 (4.64)
  Time-matched baseline (Day -1): 4-8 hours | 98.92 (8.64) | 92.27 (7.73) | 93.98 (4.94)
  Time-matched baseline (Day -1): 8-12 hours | 103.25 (8.66) | 96.20 (9.50) | 96.76 (8.22)
  Time-matched baseline (Day -1): 12-16 hours | 93.31 (9.82) | 87.07 (6.75) | 90.02 (8.80)
  Time-matched baseline (Day -1): 16-20 hours | 87.48 (10.42) | 85.54 (9.68) | 83.70 (9.24)
  Time-matched baseline (Day -1): 20-24 hours | 97.62 (11.48) | 89.30 (6.40) | 90.96 (6.46)
  Day 1, 0-4 hours | -0.40 (2.61) | -4.84 (1.86) | -5.57 (1.88)
  Day 1, 4-8 hours | 0.24 (2.86) | -4.98 (2.15) | -7.97 (2.11)
  Day 1, 8-12 hours | 0.84 (2.87) | -5.87 (2.15) | -2.30 (2.14)
  Day 1, 12-16 hours | -2.21 (1.90) | -1.84 (1.47) | -2.23 (1.44)
  Day 1, 16-20 hours | 1.47 (2.96) | -0.86 (2.28) | -0.97 (2.29)
  Day 1, 20-24 hours | 0.99 (2.20) | 0.25 (1.63) | -0.13 (1.60)
  Day 7, 0-4 hours | -2.77 (2.13) | -7.90 (1.52) | -6.41 (1.53)
  Day 7, 4-8 hours | -2.54 (2.73) | -6.46 (2.06) | -4.99 (2.02)
  Day 7, 8-12 hours | -1.71 (2.33) | -6.47 (1.74) | -2.96 (1.73)
  Day 7, 12-16 hours | -2.35 (2.42) | -4.46 (1.86) | -2.30 (1.83)
  Day 7, 16-20 hours | 2.93 (2.89) | -3.73 (2.23) | -3.45 (2.24)
  Day 7, 20-24 hours | -1.18 (2.62) | -3.47 (1.94) | -1.35 (1.91)
  Day 14, 0-4 hours: number analyzed (Participants) | 6 | 9 | 10
  Day 14, 0-4 hours | -2.65 (2.67) | -10.39 (1.99) | -6.51 (1.86)
  Day 14, 4-8 hours: number analyzed (Participants) | 6 | 9 | 10
  Day 14, 4-8 hours | -2.26 (2.38) | -11.78 (1.89) | -7.91 (1.74)
  Day 14, 8-12 hours: number analyzed (Participants) | 6 | 9 | 10
  Day 14, 8-12 hours | -1.27 (3.35) | -9.89 (2.65) | -7.32 (2.46)
  Day 14, 12-16 hours: number analyzed (Participants) | 6 | 9 | 10
  Day 14, 12-16 hours | -1.55 (3.31) | -2.91 (2.71) | -6.50 (2.49)
  Day 14, 16-20 hours: number analyzed (Participants) | 6 | 9 | 10
  Day 14, 16-20 hours | 0.05 (2.75) | -3.38 (2.23) | -5.33 (2.12)
  Day 14, 20-24 hours: number analyzed (Participants) | 6 | 9 | 10
  Day 14, 20-24 hours | -0.49 (2.70) | -0.57 (2.12) | -2.38 (1.95)
Statistical Analysis 1: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.45, 95% CI 2-sided [-11.30 to 2.41], Standard Error of Mean 3.31 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.17, 95% CI 2-sided [-12.10 to 1.75], Standard Error of Mean 3.34 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.23, 95% CI 2-sided [-12.87 to 2.42], Standard Error of Mean 3.69 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -8.22, 95% CI 2-sided [-15.64 to -0.79], Standard Error of Mean 3.58 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -6.72, 95% CI 2-sided [-14.29 to 0.86], Standard Error of Mean 3.65 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.14, 95% CI 2-sided [-10.66 to 4.38], Standard Error of Mean 3.63 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.37, 95% CI 2-sided [-4.71 to 5.45], Standard Error of Mean 2.45 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 12-16; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.02, 95% CI 2-sided [-4.94 to 4.91], Standard Error of Mean 2.37 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.33, 95% CI 2-sided [-10.07 to 5.41], Standard Error of Mean 3.73 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 10: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.45, 95% CI 2-sided [-10.26 to 5.37], Standard Error of Mean 3.77 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.75, 95% CI 2-sided [-6.62 to 5.13], Standard Error of Mean 2.83 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 12: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.13, 95% CI 2-sided [-6.83 to 4.58], Standard Error of Mean 2.75 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.13, 95% CI 2-sided [-10.72 to 0.47], Standard Error of Mean 2.70 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 14: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.64, 95% CI 2-sided [-9.29 to 2.01], Standard Error of Mean 2.72 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.92, 95% CI 2-sided [-11.22 to 3.38], Standard Error of Mean 3.52 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 16: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.46, 95% CI 2-sided [-9.54 to 4.63], Standard Error of Mean 3.42 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.75, 95% CI 2-sided [-10.90 to 1.39], Standard Error of Mean 2.96 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 18: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.25, 95% CI 2-sided [-7.35 to 4.85], Standard Error of Mean 2.94 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.11, 95% CI 2-sided [-8.57 to 4.35], Standard Error of Mean 3.11 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 20: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.05, 95% CI 2-sided [-6.21 to 6.31], Standard Error of Mean 3.02 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -6.66, 95% CI 2-sided [-14.22 to 0.90], Standard Error of Mean 3.65 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 22: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -6.38, 95% CI 2-sided [-14.01 to 1.25], Standard Error of Mean 3.68 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.29, 95% CI 2-sided [-9.30 to 4.71], Standard Error of Mean 3.38 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 24: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.17, 95% CI 2-sided [-6.97 to 6.64], Standard Error of Mean 3.28 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 25: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -7.74, 95% CI 2-sided [-15.03 to -0.44], Standard Error of Mean 3.51 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 26: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.86, 95% CI 2-sided [-10.88 to 3.16], Standard Error of Mean 3.37 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 27: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 4-8; Test type: Other — No statistical testing was performed; Least squares mean difference = -9.53, 95% CI 2-sided [-16.10 to -2.95], Standard Error of Mean 3.16 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 28: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.66, 95% CI 2-sided [-11.82 to 0.50], Standard Error of Mean 2.96 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 29: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -8.62, 95% CI 2-sided [-17.77 to 0.54], Standard Error of Mean 4.40 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 30: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -6.05, 95% CI 2-sided [-14.79 to 2.69], Standard Error of Mean 4.20 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 31: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.36, 95% CI 2-sided [-10.51 to 7.79], Standard Error of Mean 4.40 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 32: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.95, 95% CI 2-sided [-13.50 to 3.60], Standard Error of Mean 4.11 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 33: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.43, 95% CI 2-sided [-10.81 to 3.96], Standard Error of Mean 3.55 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 34: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.38, 95% CI 2-sided [-12.64 to 1.89], Standard Error of Mean 3.49 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 35: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.08, 95% CI 2-sided [-7.55 to 7.39], Standard Error of Mean 3.59 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 36: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.89, 95% CI 2-sided [-8.89 to 5.12], Standard Error of Mean 3.37 — [estimate comment as in outcome 1, analysis 2]

16. Primary Outcome: Change From Time-Matched Baseline Over Time in ABPM 24-hour Averages of Diastolic Blood Pressure
Description: as for outcome 8
Time Frame: Time Matched Baseline (Day -1), Days 1, 7, and 14
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD | IW-1973 40 mg Total Daily Dose (Overall)
Number analyzed (Participants) | 6 | 10 | 10 | 20
mmHg
  Time Matched Baseline (Day -1) | 77.37 (9.26) | 71.57 (8.58) | 71.50 (6.33) | 71.53 (7.34)
  Change at Day 1 | -1.73 (1.29) | -2.53 (0.96) | -2.82 (0.96) | -2.67 (0.69)
  Change at Day 7 | -1.60 (1.49) | -4.27 (1.12) | -3.44 (1.12) | -3.86 (0.80)
  Change at Day 14: number analyzed (Participants) | 6 | 9 | 10 | 20
  Change at Day 14 | -1.36 (2.04) | -5.33 (1.61) | -5.53 (1.51) | -5.43 (1.11)
Statistical Analysis 1: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.79, 95% CI 2-sided [-4.17 to 2.59], Standard Error of Mean 1.63 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.09, 95% CI 2-sided [-4.47 to 2.29], Standard Error of Mean 1.63 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs IW-1973 40 mg Total Daily Dose (Overall); Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.94, 95% CI 2-sided [-4.02 to 2.14], Standard Error of Mean 1.48 — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.67, 95% CI 2-sided [-6.60 to 1.26], Standard Error of Mean 1.89 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.84, 95% CI 2-sided [-5.77 to 2.10], Standard Error of Mean 1.90 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs IW-1973 40 mg Total Daily Dose (Overall); Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.25, 95% CI 2-sided [-5.83 to 1.32], Standard Error of Mean 1.72 — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.97, 95% CI 2-sided [-9.50 to 1.56], Standard Error of Mean 2.66 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.17, 95% CI 2-sided [-9.52 to 1.18], Standard Error of Mean 2.57 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs IW-1973 40 mg Total Daily Dose (Overall); Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.07, 95% CI 2-sided [-9.01 to 0.87], Standard Error of Mean 2.38 — [estimate comment as in outcome 8, analysis 1]

17. Primary Outcome: Change From Time-Matched Baseline Over Time in ABPM Daytime (12-hour) Averages of Diastolic Blood Pressure
Description: as for outcome 9
Time Frame: Time Matched Baseline (Day -1), Days 1, 7, and 14
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
mmHg
  Time Matched Baseline (Day -1) | 80.71 (8.65) | 74.31 (9.19) | 74.20 (6.45)
  Change at Day 1 | -0.88 (1.76) | -4.28 (1.31) | -4.47 (1.31)
  Change at Day 7 | -2.36 (1.61) | -5.66 (1.20) | -4.36 (1.20)
  Change at Day 14: number analyzed (Participants) | 6 | 9 | 10
  Change at Day 14 | -1.59 (2.03) | -8.88 (1.59) | -6.69 (1.50)
Statistical Analysis 1: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.40, 95% CI 2-sided [-8.01 to 1.21], Standard Error of Mean 2.22 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.60, 95% CI 2-sided [-8.21 to 1.02], Standard Error of Mean 2.23 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.30, 95% CI 2-sided [-7.53 to 0.92], Standard Error of Mean 2.04 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.01, 95% CI 2-sided [-6.24 to 2.23], Standard Error of Mean 2.04 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = -7.29, 95% CI 2-sided [-12.80 to -1.79], Standard Error of Mean 2.65 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.10, 95% CI 2-sided [-10.43 to 0.23], Standard Error of Mean 2.56 — [estimate comment as in outcome 1, analysis 2]

18. Primary Outcome: Change From Time-Matched Baseline Over Time in ABPM Nighttime (12-Hour) Averages of Diastolic Blood Pressure
Description: as for outcome 10
Time Frame: Time Matched Baseline (Day -1), Days 1, 7, and 14
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
mmHg
  Time Matched Baseline (Day -1) | 73.42 (10.04) | 68.44 (8.60) | 68.36 (6.80)
  Change at Day 1 | -2.02 (1.51) | -1.03 (1.14) | -1.46 (1.14)
  Change at Day 7 | -0.42 (1.94) | -2.96 (1.47) | -2.68 (1.47)
  Change at Day 14: number analyzed (Participants) | 6 | 9 | 10
  Change at Day 14 | -0.81 (2.41) | -1.84 (1.92) | -4.48 (1.81)
Statistical Analysis 1: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.99, 95% CI 2-sided [-2.97 to 4.95], Standard Error of Mean 1.91 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.55, 95% CI 2-sided [-3.41 to 4.52], Standard Error of Mean 1.91 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.54, 95% CI 2-sided [-7.63 to 2.56], Standard Error of Mean 2.46 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.26, 95% CI 2-sided [-7.36 to 2.85], Standard Error of Mean 2.46 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.03, 95% CI 2-sided [-7.55 to 5.49], Standard Error of Mean 3.13 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.68, 95% CI 2-sided [-10.00 to 2.65], Standard Error of Mean 3.04 — [estimate comment as in outcome 1, analysis 2]

19. Primary Outcome: Change From Time-Matched Baseline Over Time in ABPM 4-hour Averages of Diastolic Blood Pressure
Description: as for outcome 11
Time Frame: Time-matched baseline (Day -1), Days 1, 7, 14: 0-4, 4-8, 8-12, 12-16, 16-20, 20-24 hours postdose
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
mmHg
  Time Matched Baseline (Day -1): 0-4 hours | 78.96 (8.70) | 72.48 (8.58) | 71.58 (5.46)
  Time Matched Baseline (Day -1): 4-8 hours | 79.85 (9.34) | 73.96 (8.85) | 73.79 (6.71)
  Time Matched Baseline (Day -1): 8-12 hours | 83.31 (8.49) | 76.47 (11.76) | 77.13 (8.49)
  Time Matched Baseline (Day -1): 12-16 hours | 74.27 (10.88) | 68.10 (7.92) | 70.29 (8.87)
  Time Matched Baseline (Day -1): 16-20 hours | 70.07 (9.16) | 67.89 (10.04) | 64.87 (8.26)
  Time Matched Baseline (Day -1): 20-24 hours | 77.61 (10.95) | 70.57 (8.35) | 71.04 (7.34)
  Day 1, 0-4 hours | -0.57 (1.98) | -3.15 (1.45) | -4.63 (1.47)
  Day 1, 4-8 hours | -1.02 (2.15) | -4.88 (1.61) | -5.75 (1.61)
  Day 1, 8-12 hours | -0.08 (2.64) | -5.18 (1.99) | -3.04 (1.99)
  Day 1, 12-16 hours | -2.99 (2.10) | -2.12 (1.61) | -2.44 (1.59)
  Day 1, 16-20 hours | -1.41 (2.56) | -1.97 (1.96) | -1.87 (1.99)
  Day 1, 20-24 hours | -0.13 (1.89) | 1.59 (1.41) | 0.12 (1.40)
  Day 7, 0-4 hours | -1.88 (1.56) | -6.31 (1.14) | -6.05 (1.15)
  Day 7, 4-8 hours | -2.55 (2.45) | -5.94 (1.83) | -3.61 (1.84)
  Day 7, 8-12 hours | -2.16 (2.01) | -4.98 (1.52) | -3.52 (1.51)
  Day 7, 12-16 hours | -2.18 (2.32) | -3.37 (1.78) | -3.45 (1.75)
  Day 7, 16-20 hours | 2.29 (2.62) | -3.57 (2.01) | -3.91 (2.03)
  Day 7, 20-24 hours | -0.13 (2.37) | -1.74 (1.77) | -0.76 (1.76)
  Day 14, 0-4 hours | -2.02 (2.16) | -8.92 (1.66) | -6.06 (1.57)
  Day 14, 4-8 hours | -1.52 (1.98) | -9.77 (1.56) | -7.07 (1.47)
  Day 14, 8-12 hours | -0.98 (2.99) | -8.06 (2.39) | -6.83 (2.24)
  Day 14, 12-16 hours | -0.91 (3.19) | -2.32 (2.59) | -6.07 (2.40)
  Day 14, 16-20 hours | -0.94 (2.91) | -3.30 (2.34) | -5.44 (2.24)
  Day 14, 20-24 hours | 0.50 (2.64) | 0.06 (2.08) | -1.48 (1.95)
Statistical Analysis 1: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.58, 95% CI 2-sided [-7.76 to 2.59], Standard Error of Mean 2.49 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.06, 95% CI 2-sided [-9.32 to 1.19], Standard Error of Mean 2.53 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.86, 95% CI 2-sided [-9.51 to 1.80], Standard Error of Mean 2.73 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.73, 95% CI 2-sided [-10.40 to 0.93], Standard Error of Mean 2.73 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.10, 95% CI 2-sided [-12.06 to 1.86], Standard Error of Mean 3.36 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.96, 95% CI 2-sided [-9.87 to 3.96], Standard Error of Mean 3.33 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.87, 95% CI 2-sided [-4.70 to 6.45], Standard Error of Mean 2.69 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.55, 95% CI 2-sided [-4.90 to 6.01], Standard Error of Mean 2.63 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.56, 95% CI 2-sided [-7.22 to 6.10], Standard Error of Mean 3.21 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 10: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.47, 95% CI 2-sided [-7.27 to 6.34], Standard Error of Mean 3.28 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.72, 95% CI 2-sided [-3.26 to 6.69], Standard Error of Mean 2.40 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 12: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.25, 95% CI 2-sided [-4.69 to 5.20], Standard Error of Mean 2.38 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.43, 95% CI 2-sided [-8.50 to -0.36], Standard Error of Mean 1.96 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 14: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.17, 95% CI 2-sided [-8.30 to -0.03], Standard Error of Mean 1.99 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -3.39, 95% CI 2-sided [-9.82 to 3.04], Standard Error of Mean 3.10 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 16: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.06, 95% CI 2-sided [-7.51 to 5.38], Standard Error of Mean 3.11 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.82, 95% CI 2-sided [-8.12 to 2.48], Standard Error of Mean 2.56 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 18: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.36, 95% CI 2-sided [-6.63 to 3.91], Standard Error of Mean 2.54 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.19, 95% CI 2-sided [-7.35 to 4.97], Standard Error of Mean 2.97 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 20: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.26, 95% CI 2-sided [-7.30 to 4.77], Standard Error of Mean 2.91 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.86, 95% CI 2-sided [-12.68 to 0.95], Standard Error of Mean 3.29 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 22: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -6.20, 95% CI 2-sided [-13.16 to 0.76], Standard Error of Mean 3.36 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.61, 95% CI 2-sided [-7.87 to 4.65], Standard Error of Mean 3.02 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 24: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.63, 95% CI 2-sided [-6.85 to 5.59], Standard Error of Mean 3.00 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 25: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -6.91, 95% CI 2-sided [-12.74 to -1.08], Standard Error of Mean 2.80 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 26: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.04, 95% CI 2-sided [-9.73 to 1.66], Standard Error of Mean 2.74 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 27: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -8.25, 95% CI 2-sided [-13.59 to -2.91], Standard Error of Mean 2.57 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 28: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.56, 95% CI 2-sided [-10.76 to -0.35], Standard Error of Mean 2.50 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 29: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -7.07, 95% CI 2-sided [-15.20 to 1.05], Standard Error of Mean 3.91 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 30: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.85, 95% CI 2-sided [-13.68 to 1.98], Standard Error of Mean 3.77 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 31: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.40, 95% CI 2-sided [-10.14 to 7.33], Standard Error of Mean 4.20 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 32: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -5.16, 95% CI 2-sided [-13.46 to 3.14], Standard Error of Mean 3.99 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 33: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -2.37, 95% CI 2-sided [-10.14 to 5.40], Standard Error of Mean 3.74 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 34: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -4.51, 95% CI 2-sided [-12.25 to 3.23], Standard Error of Mean 3.72 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 35: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.44, 95% CI 2-sided [-7.60 to 6.72], Standard Error of Mean 3.44 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 36: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.98, 95% CI 2-sided [-8.88 to 4.92], Standard Error of Mean 3.32 — [estimate comment as in outcome 1, analysis 2]

20. Primary Outcome: Change From Time-Matched Baseline Over Time in ABPM 24-hour Averages of Pulse
Description: as for outcome 8
Time Frame: Time Matched Baseline (Day -1), Days 1, 7, and 14
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment.
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD | IW-1973 40 mg Total Daily Dose (Overall)
Number analyzed (Participants) | 6 | 10 | 10 | 20
bpm
  Time Matched Baseline (Day -1) | 75.08 (14.09) | 72.81 (10.79) | 75.40 (10.84) | 74.10 (10.61)
  Change at Day 1 | -0.90 (1.25) | 2.29 (0.97) | 2.64 (0.97) | 2.47 (0.69)
  Change at Day 7 | -1.92 (1.38) | 2.67 (1.08) | 2.57 (1.07) | 2.62 (0.76)
  Change at Day 14: number analyzed (Participants) | 6 | 9 | 10 | 20
  Change at Day 14 | -0.45 (1.50) | 2.12 (1.23) | 2.71 (1.16) | 2.42 (0.84)
Statistical Analysis 1: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = 3.19, 95% CI 2-sided [-0.10 to 6.48], Standard Error of Mean 1.59 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = 3.53, 95% CI 2-sided [0.25 to 6.82], Standard Error of Mean 1.58 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs IW-1973 40 mg Total Daily Dose (Overall); Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = 3.36, 95% CI 2-sided [0.40 to 6.32], Standard Error of Mean 1.43 — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = 4.59, 95% CI 2-sided [0.95 to 8.23], Standard Error of Mean 1.76 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = 4.49, 95% CI 2-sided [0.86 to 8.12], Standard Error of Mean 1.75 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs IW-1973 40 mg Total Daily Dose (Overall); Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = 4.54, 95% CI 2-sided [1.27 to 7.81], Standard Error of Mean 1.58 — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = 2.58, 95% CI 2-sided [-1.45 to 6.61], Standard Error of Mean 1.94 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = 3.17, 95% CI 2-sided [-0.78 to 7.11], Standard Error of Mean 1.90 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs IW-1973 40 mg Total Daily Dose (Overall); Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = 2.87, 95% CI 2-sided [-0.71 to 6.45], Standard Error of Mean 1.72 — [estimate comment as in outcome 8, analysis 1]

21. Primary Outcome: Change From Time-Matched Baseline Over Time in ABPM Daytime (12-hour) Averages of Pulse
Description: as for outcome 9
Time Frame: Time Matched Baseline (Day -1), Days 1, 7, and 14
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment.
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
bpm
  Time Matched Baseline (Day -1) | 76.81 (15.00) | 75.98 (12.84) | 78.18 (11.47)
  Change at Day 1 | 0.14 (1.84) | 2.30 (1.42) | 4.23 (1.43)
  Change at Day 7 | -1.80 (1.51) | 2.75 (1.17) | 2.22 (1.17)
  Change at Day 14: number analyzed (Participants) | 6 | 9 | 10
  Change at Day 14 | -0.46 (1.59) | 2.66 (1.30) | 3.28 (1.23)
Statistical Analysis 1: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = 2.17, 95% CI 2-sided [-2.65 to 6.99], Standard Error of Mean 2.32 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = 4.09, 95% CI 2-sided [-0.73 to 8.91], Standard Error of Mean 2.33 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = 4.56, 95% CI 2-sided [0.60 to 8.51], Standard Error of Mean 1.91 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = 4.02, 95% CI 2-sided [0.07 to 7.98], Standard Error of Mean 1.91 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = 3.12, 95% CI 2-sided [-1.15 to 7.39], Standard Error of Mean 2.05 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = 3.74, 95% CI 2-sided [-0.44 to 7.92], Standard Error of Mean 2.01 — [estimate comment as in outcome 1, analysis 2]

22. Primary Outcome: Change From Time-Matched Baseline Over Time in ABPM Nighttime (12-Hour) Averages of Pulse
Description: as for outcome 10
Time Frame: Time Matched Baseline (Day -1), Days 1, 7, and 14
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment.
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
bpm
  Time Matched Baseline (Day -1) | 73.43 (13.39) | 69.62 (8.91) | 72.54 (10.46)
  Change at Day 1 | -2.01 (1.21) | 2.29 (0.94) | 0.93 (0.94)
  Change at Day 7 | -2.24 (1.63) | 2.57 (1.27) | 2.86 (1.26)
  Change at Day 14: number analyzed (Participants) | 6 | 9 | 10
  Change at Day 14 | -0.40 (1.79) | 1.48 (1.46) | 2.15 (1.38)
Statistical Analysis 1: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = 4.30, 95% CI 2-sided [1.10 to 7.49], Standard Error of Mean 1.54 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1; Test type: Other — No statistical testing was performed; Least squares mean difference = 2.94, 95% CI 2-sided [-0.23 to 6.10], Standard Error of Mean 1.53 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = 4.80, 95% CI 2-sided [0.50 to 9.11], Standard Error of Mean 2.07 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7; Test type: Other — No statistical testing was performed; Least squares mean difference = 5.10, 95% CI 2-sided [0.84 to 9.36], Standard Error of Mean 2.05 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.89, 95% CI 2-sided [-2.93 to 6.70], Standard Error of Mean 2.32 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14; Test type: Other — No statistical testing was performed; Least squares mean difference = 2.55, 95% CI 2-sided [-2.15 to 7.25], Standard Error of Mean 2.26 — [estimate comment as in outcome 1, analysis 2]

23. Primary Outcome: Change From Time-Matched Baseline Over Time in ABPM 4-hour Averages of Pulse
Description: as for outcome 11
Time Frame: Time-matched baseline (Day -1), Days 1, 7, 14: 0-4, 4-8, 8-12, 12-16, 16-20, 20-24 hours postdose
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment.
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
bpm
  Time Matched Baseline (Day -1): 0-4 hours | 73.52 (14.02) | 73.89 (12.23) | 76.46 (9.48)
  Time Matched Baseline (Day -1): 4-8 hours | 77.65 (15.57) | 76.88 (15.09) | 79.91 (14.33)
  Time Matched Baseline (Day -1): 8-12 hours | 79.00 (15.50) | 77.34 (11.42) | 78.21 (11.67)
  Time Matched Baseline (Day -1): 12-16 hours | 78.60 (15.22) | 72.93 (9.38) | 75.36 (11.89)
  Time Matched Baseline (Day -1): 16-20 hours | 72.08 (13.37) | 67.79 (8.80) | 70.51 (10.23)
  Time Matched Baseline (Day -1): 20-24 hours | 68.05 (11.26) | 67.97 (8.75) | 71.45 (10.35)
  Day 1, 0-4 hours | 0.87 (2.07) | 7.68 (1.60) | 7.42 (1.60)
  Day 1, 4-8 hours | 1.18 (2.76) | 0.23 (2.14) | 3.02 (2.14)
  Day 1, 8-12 hours | -0.96 (2.14) | -1.33 (1.65) | 2.15 (1.65)
  Day 1, 12-16 hours | -4.33 (1.68) | 2.13 (1.30) | 1.24 (1.29)
  Day 1, 16-20 hours | -1.67 (1.24) | 1.95 (0.97) | 0.73 (0.96)
  Day 1, 20-24 hours | 0.76 (1.77) | 2.50 (1.37) | 1.09 (1.38)
  Day 7, 0-4 hours | -0.09 (2.11) | 4.27 (1.63) | 5.32 (1.64)
  Day 7, 4-8 hours | -2.94 (1.72) | 1.95 (1.34) | 1.36 (1.34)
  Day 7, 8-12 hours | -2.25 (1.78) | 1.79 (1.38) | 0.01 (1.38)
  Day 7, 12-16 hours | -4.05 (1.89) | 2.85 (1.46) | 2.10 (1.45)
  Day 7, 16-20 hours | -2.56 (1.87) | 2.44 (1.45) | 2.78 (1.44)
  Day 7, 20-24 hours | 0.23 (1.85) | 1.91 (1.44) | 4.26 (1.44)
  Day 14, 0-4 hours: number analyzed (Participants) | 6 | 9 | 10
  Day 14, 0-4 hours | 0.77 (1.95) | 4.82 (1.59) | 4.53 (1.51)
  Day 14, 4-8 hours: number analyzed (Participants) | 6 | 9 | 10
  Day 14, 4-8 hours | -2.85 (2.56) | 2.33 (2.09) | 2.76 (1.99)
  Day 14, 8-12 hours: number analyzed (Participants) | 6 | 9 | 10
  Day 14, 8-12 hours | 0.89 (1.91) | 0.68 (1.56) | 2.50 (1.48)
  Day 14, 12-16 hours: number analyzed (Participants) | 6 | 9 | 10
  Day 14, 12-16 hours | -3.74 (2.33) | 1.35 (1.89) | 1.56 (1.79)
  Day 14, 16-20 hours: number analyzed (Participants) | 6 | 9 | 10
  Day 14, 16-20 hours | -0.88 (1.98) | 0.43 (1.61) | 2.06 (1.53)
  Day 14, 20-24 hours: number analyzed (Participants) | 6 | 9 | 10
  Day 14, 20-24 hours | 4.14 (2.31) | 2.80 (1.88) | 3.00 (1.80)
Statistical Analysis 1: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 6.81, 95% CI 2-sided [1.40 to 12.22], Standard Error of Mean 2.61 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 6.55, 95% CI 2-sided [1.12 to 11.99], Standard Error of Mean 2.62 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.95, 95% CI 2-sided [-8.18 to 6.28], Standard Error of Mean 3.49 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.85, 95% CI 2-sided [-5.39 to 9.09], Standard Error of Mean 3.49 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.38, 95% CI 2-sided [-5.98 to 5.23], Standard Error of Mean 2.70 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 3.10, 95% CI 2-sided [-2.50 to 8.70], Standard Error of Mean 2.70 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 6.46, 95% CI 2-sided [2.02 to 10.89], Standard Error of Mean 2.14 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 5.57, 95% CI 2-sided [1.19 to 9.95], Standard Error of Mean 2.11 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 3.63, 95% CI 2-sided [0.34 to 6.91], Standard Error of Mean 1.59 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 10: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 2.41, 95% CI 2-sided [-0.84 to 5.66], Standard Error of Mean 1.57 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 1, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.74, 95% CI 2-sided [-2.89 to 6.36], Standard Error of Mean 2.23 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 12: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 1, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 0.33, 95% CI 2-sided [-4.33 to 4.99], Standard Error of Mean 2.25 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 4.36, 95% CI 2-sided [-1.17 to 9.88], Standard Error of Mean 2.66 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 14: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 5.41, 95% CI 2-sided [-0.14 to 10.96], Standard Error of Mean 2.68 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 4.88, 95% CI 2-sided [0.36 to 9.40], Standard Error of Mean 2.18 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 16: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 4.30, 95% CI 2-sided [-0.22 to 8.83], Standard Error of Mean 2.18 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 4.04, 95% CI 2-sided [-0.65 to 8.72], Standard Error of Mean 2.26 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 18: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 2.26, 95% CI 2-sided [-2.42 to 6.94], Standard Error of Mean 2.26 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 6.90, 95% CI 2-sided [1.91 to 11.89], Standard Error of Mean 2.41 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 20: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 6.15, 95% CI 2-sided [1.22 to 11.08], Standard Error of Mean 2.38 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 4.99, 95% CI 2-sided [0.05 to 9.93], Standard Error of Mean 2.38 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 22: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 5.34, 95% CI 2-sided [0.45 to 10.22], Standard Error of Mean 2.36 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 7, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.67, 95% CI 2-sided [-3.17 to 6.52], Standard Error of Mean 2.33 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 24: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 7, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 4.03, 95% CI 2-sided [-0.86 to 8.92], Standard Error of Mean 2.36 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 25: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 4.05, 95% CI 2-sided [-1.18 to 9.27], Standard Error of Mean 2.51 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 26: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 0-4 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 3.76, 95% CI 2-sided [-1.38 to 8.90], Standard Error of Mean 2.47 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 27: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 5.18, 95% CI 2-sided [-1.70 to 12.06], Standard Error of Mean 3.31 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 28: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 4-8 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 5.61, 95% CI 2-sided [-1.14 to 12.37], Standard Error of Mean 3.25 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 29: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.21, 95% CI 2-sided [-5.35 to 4.92], Standard Error of Mean 2.47 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 30: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 8-12 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.61, 95% CI 2-sided [-3.42 to 6.65], Standard Error of Mean 2.42 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 31: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 5.08, 95% CI 2-sided [-1.19 to 11.36], Standard Error of Mean 3.02 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 32: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 12-16 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 5.30, 95% CI 2-sided [-0.83 to 11.42], Standard Error of Mean 2.94 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 33: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 14, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 1.30, 95% CI 2-sided [-4.02 to 6.63], Standard Error of Mean 2.56 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 34: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 16-20 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = 2.93, 95% CI 2-sided [-2.26 to 8.12], Standard Error of Mean 2.50 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 35: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.34, 95% CI 2-sided [-7.52 to 4.85], Standard Error of Mean 2.98 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 36: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 14, 20-24 hours; Test type: Other — No statistical testing was performed; Least squares mean difference = -1.14, 95% CI 2-sided [-7.25 to 4.98], Standard Error of Mean 2.94 — [estimate comment as in outcome 1, analysis 2]

24. Primary Outcome: Change From Baseline in Reactive Hyperemia Index (RHI) on Day 13
Description: RHI is a measure of the extent of vessel dilatation and augmentation in vascular blood flow after a prespecified period of flow interruption. RHI is determined as the ratio of the post-to-pre- occlusion peripheral arterial tonometry amplitude of the tested (occluded) arm, divided by the post to-pre-occlusion ratio of the control arm. RHI values >1.67 indicate normal endothelial function, while values ≤1.67 indicate endothelial dysfunction.
Time Frame: Baseline, Day 13 predose AM
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment. Participants with an assessment.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD | IW-1973 40 mg Total Daily Dose (Overall)
Number analyzed (Participants) | 6 | 10 | 9 | 19
ratio
  Baseline | 2.327 (1.118) | 1.918 (0.587) | 1.683 (0.379) | 1.807 (0.501)
  Day 13 predose AM | 0.282 (0.219) | -0.006 (0.163) | 0.177 (0.176) | 0.086 (0.120)
Statistical Analysis 1: Comparison: Placebo vs IW-1973 40 mg BID/QD; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.288, 95% CI 2-sided [-0.857 to 0.282], Standard Error of Mean 0.274 — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs IW-1973 40 mg QD/QD; Test type: Other — No statistical testing was performed; Least squares mean difference = -0.105, 95% CI 2-sided [-0.708 to 0.498], Standard Error of Mean 0.290 — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs IW-1973 40 mg Total Daily Dose (Overall); Test type: Other — No statistical testing was performed; Least squares mean difference = -0.196, 95% CI 2-sided [-0.727 to 0.335], Standard Error of Mean 0.255 — [estimate comment as in outcome 8, analysis 1]

25. Primary Outcome: Post-Baseline Platelet Reactivity on Days 8 and 14: P2Y12 Reaction Units (PRU) Assay
Description: Platelet reactivity, as measured by VerifyNow PRU assay, and presented as number of participants with < 180 PRU or ≥ 180 PRU post-baseline (Days 8 and 14), by baseline category.
  The VerifyNow PRU assay measures effects on platelet activation caused by inhibition of the platelet receptor, P2Y12. This receptor is activated by adenosine 5'-diphosphate (ADP) in the cascade leading to platelet aggregation but can be blocked by P2Y12 inhibitor drugs, such as clopidogrel. Blockage of this receptor diminishes platelet activation and the ability of platelets to bind to fibrinogen. VerifyNow PRU assay values < 180 units indicate impairment of platelet aggregation.
Time Frame: Baseline, Day 8, Day 14
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment. Participants with a baseline (BL) and postbaseline (PBL) assessment at given time point, by specific BL category < 180 or ≥ 180 PRU.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 5 | 10 | 10
Participants
  Baseline: <180 PRU | 0 | 0 | 0
  Baseline: ≥180 PRU | 5 | 10 | 10
  PRU Day 8: <180 BL, <180 PBL: number analyzed (Participants) | 0 | 0 | 0
  PRU Day 8: <180 BL, ≥180 PBL: number analyzed (Participants) | 0 | 0 | 0
  PRU Day 8: ≥180 BL, <180 PBL | 0 | 0 | 0
  PRU Day 8: ≥180 BL, ≥180 PBL | 5 | 10 | 10
  PRU Day 14: <180 BL, <180 PBL: number analyzed (Participants) | 0 | 0 | 0
  PRU Day 14: <180 BL, ≥180 PBL: number analyzed (Participants) | 0 | 0 | 0
  PRU Day 14: ≥180 BL, <180 PBL | 0 | 0 | 0
  PRU Day 14: ≥180 BL, ≥180 PBL | 5 | 10 | 10

26. Primary Outcome: Post-Baseline Platelet Reactivity on Days 8 and 14: Aspirin Reaction Units (ARU) Assay
Description: Platelet reactivity, as measured by VerifyNow ARU assay, and presented as number of participants with ≤ 549 ARU or > 549 ARU post-baseline (Days 8 and 14), by baseline category.
  Aspirin irreversibly inhibits cyclooxygenase 1, which converts arachidonic acid to thromboxane A2, which in turn is involved in the activation of the glycoprotein (GP)IIb/IIIa receptor necessary to initiate platelet aggregation. Impairment of platelet aggregation of the aspirin type is defined for the VerifyNow aspirin assay as values ≤ 549 ARU.
Time Frame: Baseline, Day 8, Day 14
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment. Participants with a baseline (BL) and postbaseline (PBL) assessment at given time point, by specific BL category (≤ 549 or > 549 ARU).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 5 | 10 | 10
Participants
  Baseline: ≤ 549 ARU | 2 | 5 | 6
  Baseline: > 549 ARU | 3 | 5 | 4
  Day 8: ≤ 549 BL, ≤ 549 PBL: number analyzed (Participants) | 2 | 5 | 6
  Day 8: ≤ 549 BL, ≤ 549 PBL | 2 | 5 | 6
  Day 8: ≤ 549 BL, > 549 PBL: number analyzed (Participants) | 2 | 5 | 6
  Day 8: ≤ 549 BL, > 549 PBL | 0 | 0 | 0
  Day 8: > 549 BL, ≤ 549 PBL: number analyzed (Participants) | 3 | 5 | 4
  Day 8: > 549 BL, ≤ 549 PBL | 1 | 2 | 0
  Day 8: > 549 BL, > 549 PBL: number analyzed (Participants) | 3 | 5 | 4
  Day 8: > 549 BL, > 549 PBL | 2 | 3 | 4
  Day 14: ≤ 549 BL, ≤ 549 PBL: number analyzed (Participants) | 2 | 5 | 6
  Day 14: ≤ 549 BL, ≤ 549 PBL | 2 | 2 | 6
  Day 14: ≤ 549 BL, > 549 PBL: number analyzed (Participants) | 2 | 5 | 6
  Day 14: ≤ 549 BL, > 549 PBL | 0 | 3 | 0
  Day 14: > 549 BL, ≤ 549 PBL: number analyzed (Participants) | 3 | 5 | 4
  Day 14: > 549 BL, ≤ 549 PBL | 0 | 0 | 1
  Day 14: > 549 BL, > 549 PBL: number analyzed (Participants) | 3 | 5 | 4
  Day 14: > 549 BL, > 549 PBL | 3 | 5 | 3

27. Primary Outcome: Change From Study Baseline Over Time in Platelet Function Assessments: PRU Assay
Description: The VerifyNow PRU assay measures effects on platelet activation caused by inhibition of the platelet receptor, P2Y12. This receptor is activated by adenosine 5'-diphosphate (ADP) in the cascade leading to platelet aggregation but can be blocked by P2Y12 inhibitor drugs, such as clopidogrel. Blockage of this receptor diminishes platelet activation and the ability of platelets to bind to fibrinogen. VerifyNow PRU assay values <180 PRU indicate impairment of platelet aggregation.
Time Frame: Study Baseline (Day 1 predose), Day 8 (predose AM), Day 14 (predose AM)
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment. Participants with a baseline (BL) and postbaseline (PBL) assessment at given time point.
Measure: Mean (Standard Deviation); unit: PRU
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 5 | 10 | 10
PRU
  Study Baseline (Day 1 predose) | 304.0 (48.8) | 283.6 (43.1) | 294.4 (36.9)
  Change at Day 8 | -9.4 (47.8) | 8.2 (31.4) | -0.7 (36.4)
  Change at Day 14 | -4.4 (38.1) | 24.4 (38.2) | 8.5 (24.5)

28. Primary Outcome: Change From Study Baseline Over Time in Platelet Function Assessments: ARU Assay
Description: Aspirin irreversibly inhibits cyclooxygenase 1, which converts arachidonic acid to thromboxane A2, which in turn is involved in the activation of the GPIIb IIIa receptor necessary to initiate platelet aggregation. Impairment of platelet aggregation of the aspirin type is defined for the VerifyNow aspirin assay as values ≤ 549 ARU.
Time Frame: Study Baseline (Day 1 predose), Day 8 (pre AM dose), Day 14 (pre AM dose)
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: ARU
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 5 | 10 | 10
ARU
  Study Baseline (Day 1 predose) | 571.4 (82.5) | 557.4 (76.3) | 524.6 (89.5)
  Change at Day 8 | -8.0 (58.5) | -16.2 (50.9) | 18.7 (29.4)
  Change at Day 14 | 10.2 (19.8) | 30.2 (34.9) | -11.7 (34.9)

29. Primary Outcome: Percent Change From Study Baseline Over Time in HOMA-IR in Participants Without Concomitant Use of Insulin
Description: Blood samples were taken for fasting glucose and insulin levels. From these results, insulin resistance was then estimated using the updated homeostasis model assessment method for insulin resistance (HOMA-IR) computer algorithm. A higher HOMA-IR indicates a higher degree of insulin resistance. Typically a cutoff of HOMA-IR for identifying those with insulin resistance is 2.5.
Time Frame: Study baseline (defined as the last non-missing assessment before the first administration of study drug), Day 8, pre-AM dose, Day 15
Population: PD Population: all participants who received at least 1 dose of study drug and had at least 1 postdose PD assessment. Participants with a baseline (BL) and postbaseline (PBL) assessment at given time point who did not use concomitant insulin.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD | IW-1973 40 mg Total Daily Dose (Overall)
Number analyzed (Participants) | 4 | 5 | 7 | 12
percent change
  Study Baseline (Day 1 predose) | 7.350 (5.236) | 6.646 (3.403) | 7.187 (5.684) | 6.962 (4.681)
  Day 8 | -4.284 (20.823) | -27.473 (18.639) | -18.318 (15.735) | -22.895 (12.191)
  Day 15: number analyzed (Participants) | 4 | 5 | 6 | 11
  Day 15 | -12.839 (12.565) | -38.228 (11.263) | -34.015 (10.270) | -36.121 (7.609)
Statistical Analysis 1: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 8; Test type: Other — No statistical testing was performed; Least squares mean difference = -23.188, 95% CI 2-sided [-84.130 to 37.753], Standard Error of Mean 27.970 — Least Squares mean difference and associated 95% confidence interval (CI) is from an analysis of covariance (ANCOVA) model with treatment as fixed effect and baseline as covariate. Standard Error of the Mean=Standard Error of the LS Mean Difference
Statistical Analysis 2: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 8; Test type: Other — No statistical testing was performed; Least squares mean difference = -14.033, 95% CI 2-sided [-70.883 to 42.817], Standard Error of Mean 26.092 — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs IW-1973 40 mg Total Daily Dose (Overall); Day 8; Test type: Other — No statistical testing was performed; Least squares mean difference = -18.611, 95% CI 2-sided [-71.204 to 33.982], Standard Error of Mean 24.138 — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs IW-1973 40 mg BID/QD; Day 15; Test type: Other — No statistical testing was performed; Least squares mean difference = -25.389, 95% CI 2-sided [-62.551 to 11.774], Standard Error of Mean 16.885 — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs IW-1973 40 mg QD/QD; Day 15; Test type: Other — No statistical testing was performed; Least squares mean difference = -21.176, 95% CI 2-sided [-56.879 to 14.527], Standard Error of Mean 16.221 — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs IW-1973 40 mg Total Daily Dose (Overall); Day 15; Test type: Other — No statistical testing was performed; Least squares mean difference = -23.282, 95% CI 2-sided [-55.618 to 9.053], Standard Error of Mean 14.691 — [estimate comment as in outcome 29, analysis 1]

30. Primary Outcome: IW-1973 Pharmacokinetics: Area Under the Plasma Concentration Time Curve During a Dosing Interval (AUCtau) on Days 1 and 7
Description: Equivalent to AUC from time 0 to the last measurable concentration (AUClast), with time of last measurable concentration (Tlast)=12 hours for BID dosing and Tlast=24 hours for QD dosing.
Time Frame: Days 1 and 7 (AM): 1, 3, and 6 hours postdose
Population: Pharmacokinetic (PK) Population: all participants who received ≥1 dose of IW-1973 and had ≥1 postdose PK parameter assessment without events or deviations affecting the PK results.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- IW-1973 40 mg BID/QD: 20 mg AM; IW-1973 40 mg BID/QD: 20 mg PM: IW-1973 20 mg oral tablet taken in AM and 20 mg oral tablet taken in PM on Days 1-7.
  IW-1973 40 mg oral tablet taken QD in AM and placebo oral tablet taken QD in PM on Days 8-14.
- IW-1973 40 mg QD/QD: 40 mg AM: IW-1973 40 mg oral tablet taken QD in AM and placebo taken QD in PM on Days 1-14.
Arm/Group | IW-1973 40 mg BID/QD: 20 mg AM | IW-1973 40 mg BID/QD: 20 mg PM | IW-1973 40 mg QD/QD: 40 mg AM
Number analyzed (Participants) | 10 | 10 | 10
h*ng/mL
  Day 1 | 362 (88) | 339 (134) | 1190 (499)
  Day 7: number analyzed (Participants) | 10 | 0 | 10
  Day 7 | 795 (186) |  | 2200 (591)

31. Primary Outcome: IW-1973 Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax) on Days 1 and 7
Time Frame: Days 1 and 7 (AM): 1, 3, and 6 hours postdose
Population: PK Population: all participants who received ≥1 dose of IW-1973 and had ≥1 postdose PK parameter assessment without events or deviations affecting the PK results.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | IW-1973 40 mg BID/QD: 20 mg AM | IW-1973 40 mg BID/QD: 20 mg PM | IW-1973 40 mg QD/QD: 40 mg AM
Number analyzed (Participants) | 10 | 10 | 10
ng/mL
  Day 1 | 73.8 (18.9) | 47.8 (22.2) | 181 (107)
  Day 7: number analyzed (Participants) | 10 | 0 | 10
  Day 7 | 117 (32.6) |  | 242 (80.0)

32. Primary Outcome: IW-1973 Pharmacokinetics: Time to Cmax on Days 1 and 7
Time Frame: Days 1 and 7 (AM): 1, 3, and 6 hours postdose
Population: as for outcome 31
Measure: Median (Full Range); unit: hours
Arm/Group | IW-1973 40 mg BID/QD: 20 mg AM | IW-1973 40 mg BID/QD: 20 mg PM | IW-1973 40 mg QD/QD: 40 mg AM
Number analyzed (Participants) | 10 | 10 | 10
hours
  Day 1 | 1.0 [1.0 to 3.0] | 3.0 [3.0 to 11.9] | 2.0 [1.0 to 6.0]
  Day 7: number analyzed (Participants) | 10 | 0 | 10
  Day 7 | 1.0 [1.0 to 3.0] |  | 1.0 [1.0 to 6.0]

33. Primary Outcome: IW-1973 Pharmacokinetics: Trough Plasma Concentrations at the End of the Dosing Interval (Ctrough) on Days 1, 2, 6, 7
Time Frame: Days 1 and 7: predose; Day 2 (BID AM): predose; Day 6 (BID PM/QD): predose
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | IW-1973 40 mg BID/QD: 20 mg AM | IW-1973 40 mg BID/QD: 20 mg PM | IW-1973 40 mg QD/QD: 40 mg AM
Number analyzed (Participants) | 10 | 10 | 10
ng/mL
  Day 1 | 11.6 (4.29) | 19.6 (5.04) | 15.6 (5.24)
  Day 2: number analyzed (Participants) | 10 | 0 | 0
  Day 2 | 21.0 (5.97) |  |
  Day 6: number analyzed (Participants) | 0 | 10 | 10
  Day 6 |  | 48.4 (10.1) | 53.7 (14.5)
  Day 7 | 45.6 (14.5) | 52.4 (12.8) | 57.2 (14.9)

34. Primary Outcome: IW-1973 Pharmacokinetics: Area Under the Plasma Concentration Time Curve From Time Zero to the Last Measurable Plasma Concentration (AUClast) on Days 8 and 14
Time Frame: Day 8 and 14: 1, 3, 6h (± 5 min) postdose
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: h*mg/mL
Groups:
- IW-1973 40 mg BID/QD: 40 mg AM: IW-1973 40 mg oral tablet taken QD in AM and placebo oral tablet taken QD in PM on Days 8-14.
Arm/Group | IW-1973 40 mg BID/QD: 40 mg AM | IW-1973 40 mg QD/QD: 40 mg AM
Number analyzed (Participants) | 10 | 10
h*mg/mL
  Day 8 | 1210 (264) | 1540 (482)
  Day 14 | 17100 (6980) | 23600 (8950)

35. Primary Outcome: IW-1973 Pharmacokinetics: AUCtau on Day 14
Time Frame: Day 14: 1, 3, 6h (± 5 min) postdose
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | IW-1973 40 mg BID/QD: 40 mg AM | IW-1973 40 mg QD/QD: 40 mg AM
Number analyzed (Participants) | 10 | 10
ng/mL | 2080 (442) | 2910 (770)

36. Primary Outcome: IW-1973 Pharmacokinetics: Tmax on Days 8 and 14
Time Frame: Day 8 and 14: 1, 3, 6h (± 5 min) postdose
Population: as for outcome 31
Measure: Median (Full Range); unit: hours
Arm/Group | IW-1973 40 mg BID/QD: 40 mg AM | IW-1973 40 mg QD/QD: 40 mg AM
Number analyzed (Participants) | 10 | 10
hours
  Day 8 | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 6.2]
  Day 14 | 1.0 [1.0 to 3.0] | 3.0 [1.0 to 6.0]

37. Primary Outcome: IW-1973 Pharmacokinetics: Cmax on Days 8 and 14
Time Frame: Day 8 and 14: 1, 3, 6h (± 5 min) postdose
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | IW-1973 40 mg BID/QD: 40 mg AM | IW-1973 40 mg QD/QD: 40 mg AM
Number analyzed (Participants) | 10 | 10
ng/mL
  Day 8 | 198 (56.8) | 229 (90.6)
  Day 14 | 181 (46.8) | 250 (139)

38. Primary Outcome: IW-1973 Pharmacokinetics: Ctrough on Days 13 and 14
Time Frame: Days 13 and 14: predose
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | IW-1973 40 mg BID/QD: 40 mg AM | IW-1973 40 mg QD/QD: 40 mg AM
Number analyzed (Participants) | 10 | 10
ng/mL
  Day 13 | 56.8 (19.5) | 82.4 (22.7)
  Day 14 | 65.7 (23.0) | 90.7 (26.2)

39. Primary Outcome: IW-1973 Pharmacokinetics: Apparent Total Body Clearance (CL/F) on Day 14
Time Frame: Day 14: 1, 3, 6h (± 5 min) postdose
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | IW-1973 40 mg BID/QD: 40 mg AM | IW-1973 40 mg QD/QD: 40 mg AM
Number analyzed (Participants) | 10 | 10
L/h | 20.0 (4.34) | 14.7 (3.89)

40. Primary Outcome: IW-1973 Pharmacokinetics: Apparent Volume of Distribution During the Terminal Phase (Vz/F) on Day 14
Time Frame: Day 14: 1, 3, 6h (± 5 min) postdose
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: L
Arm/Group | IW-1973 40 mg BID/QD: 40 mg AM | IW-1973 40 mg QD/QD: 40 mg AM
Number analyzed (Participants) | 10 | 10
L | 5570 (1530) | 3880 (1370)

41. Primary Outcome: IW-1973 Pharmacokinetics: Apparent Terminal Elimination Phase Half-Life (t1/2)
Time Frame: Day 14 (final dose) time points 12 hours, 24 hours, 7 days after final dose (Day 21), and 28 days after final dose(Day 42)
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | IW-1973 40 mg BID/QD: 40 mg AM | IW-1973 40 mg QD/QD: 40 mg AM
Number analyzed (Participants) | 10 | 10
hours | 197 (57.4) | 183 (43.4)

42. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Discontinuations Due to TEAEs
Description: An adverse event (AE) is any untoward medical occurrence, which does not necessarily have to have a causal relationship with study treatment. An SAE is defined as any AE occurring at any dose that results in any of the following outcomes: death; life-threatening; hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect; important medical events. TEAEs are defined as those AEs that started or worsened in severity after the initiation of study drug administration. AEs of clinical interest (AECI) included those related to bleeding and to hypotension. Study drug causality as assessed by the Investigator who was blinded to study drug assignment.
Time Frame: From first dose of study drug to End of Trial Visit (42 [± 3] days)
Population: Safety Population: participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
participants
  TEAE | 5 | 6 | 8
  SAE | 0 | 1 | 0
  Severe TEAE | 0 | 1 | 0
  Moderate TEAE | 0 | 0 | 0
  Mild TEAE | 5 | 6 | 8
  TEAE Considered Study Drug Related | 1 | 3 | 6
  TEAE Considered Not Study Drug Related | 4 | 6 | 7
  TEAE Resulting in Study Discontinuation | 0 | 1 | 0
  TEAE Resulting in Death | 0 | 0 | 0
  AECI Related to Bleeding | 0 | 1 | 0
  AECI Related to Hypotension | 1 | 1 | 0

43. Primary Outcome: Number of Participants With Clinically Meaningful Postbaseline Laboratory Test Results
Time Frame: From first dose of study drug to End of Trial Visit (42 [± 3] days)
Population: Safety Population: participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
participants | 0 | 1 | 1

44. Primary Outcome: Number of Participants With Notable Changes in Postbaseline Blood Pressure and Heart Rate Values
Description: Supine systolic blood pressure (SSBP): ≥ 180 mmHg and increase (↑) from baseline (BL) ≥ 30 mmHg; ≤ 90 mmHg and decrease (↓) from BL ≥ 30 mmHg.
  Supine diastolic blood pressure (SDBP): ≥ 105 mmHg and ↑ from BL ≥ 20 mmHg; ≤ 50 mmHg and ↓ from BL ≥ 20 mmHg.
  Supine heart rate (SHR): ≥ 110 bpm and ↑ from BL ≥ 20 bpm; ≤ 50 bpm and ↓ from BL ≥ 20 bpm.
  Standing systolic blood pressure (StSBP): ≥ 180 mmHg and increase (↑) from baseline (BL) ≥ 30 mmHg; ≤ 90 mmHg and decrease (↓) from BL ≥ 30 mmHg.
  Standing Diastolic Blood Pressure (StDBP): ≥ 105 mmHg and ↑ from BL ≥ 20 mmHg; ≤ 50 mmHg and ↓ from BL ≥ 20 mmHg.
  Standing heart rate (StHR): ≥ 110 bpm and ↑ from BL ≥ 20 bpm; ≤ 50 bpm and ↓ from BL ≥ 20 bpm.
  Orthostatic systolic blood pressure (SBP): ↓ > 20 mmHg from supine to standing.
  Orthostatic diastolic blood pressure (DBP): ↓ > 15 mmHg from supine to standing.
  Orthostatic HR: ↓ > 30 bpm from supine to standing.
Time Frame: From first dose of study drug to End of Trial Visit (42 [± 3] days)
Population: Safety Population: participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
participants
  SSBP: ≥ 180 mmHg and ↑ from BL ≥ 30 mmHg | 0 | 0 | 0
  SSBP: ≤ 90 mmHg and ↓ from BL ≥ 30 mmHg | 0 | 1 | 0
  SDBP: ≥ 105 mmHg and ↑ from BL ≥ 20 mmHg | 0 | 0 | 0
  SDBP: ≤ 50 mmHg and ↓ from BL ≥ 20 mmHg | 0 | 2 | 0
  SHR: ≥ 110 bpm and ↑ from BL ≥ 20 bpm | 1 | 2 | 0
  SHR: ≤ 50 bpm and ↓ from BL ≥ 20 bpm | 1 | 0 | 0
  StSBP: ≥ 180 mmHg and ↑ from BL ≥ 30 mmHg | 0 | 0 | 0
  StSBP: ≤ 90 mmHg and ↓ from BL ≥ 30 mmHg | 0 | 2 | 0
  StDBP: ≥ 105 mmHg and ↑ from BL ≥ 20 mmHg | 0 | 0 | 0
  StDBP: ≤ 50 mmHg and ↓ from BL ≥ 20 mmHg | 0 | 1 | 0
  StHR: ≥ 120 bpm and ↑ from BL ≥ 25 bpm | 0 | 1 | 1
  StHR: ≤ 50 bpm and ↓ from BL ≥ 20 bpm | 0 | 0 | 0
  Orthostatic SBP: ↓ > 20 mmHg, Supine to Standing | 2 | 4 | 3
  Orthostatic DBP: ↓ > 15 mmHg, Supine to Standing | 1 | 1 | 0
  Orthostatic HR: ↑ > 30 bpm, Supine to Standing | 2 | 2 | 1

45. Primary Outcome: Number of Participants With Clinically Significant Post-Randomization Physical Examination Findings
Description: Physical examinations included examination and assessment of the following: general appearance, lymph nodes, skin, cardiovascular system, head, eyes, ears, nose, and throat, central nervous system, respiratory system, neck, peripheral nervous system, abdomen/liver/spleen, musculoskeletal system.
Time Frame: Post-randomization to End of Trial Visit (42 [± 3] days)
Population: Safety Population: participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
participants | 0 | 0 | 0

46. Primary Outcome: Number of Participants With Clinically Significant Postbaseline 12-Lead Electrocardiogram (ECG) Results
Time Frame: From first dose of study drug to End of Trial Visit (42 [± 3] days)
Population: Safety Population: participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
participants | 0 | 0 | 0

47. Primary Outcome: Change From Study Baseline Over Time in Estimated Glomerular Filtration Rate (eGFR)
Time Frame: Study Baseline, Day 15/Discharge, Day 42/End of Trial
Population: Safety Population: participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
Number analyzed (Participants) | 6 | 10 | 10
mL/min/1.73m^2
  Study Baseline | 103.045 (7.542) | 89.014 (19.729) | 80.373 (19.716)
  Day 15/Discharge | 0.158 (4.050) | -2.232 (7.275) | 1.663 (5.803)
  Day 42/End of Trial | -3.727 (10.262) | -8.905 (4.293) | -5.587 (6.196)

ADVERSE EVENTS:
Time Frame: From first dose of study drug to End of Trial Visit (42 [± 3] days)
Arm/Group | Placebo | IW-1973 40 mg BID/QD | IW-1973 40 mg QD/QD
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 5/6 | 6/10 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | IW-1973 40 mg BID/QD (N=10) | IW-1973 40 mg QD/QD (N=10)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | IW-1973 40 mg BID/QD (N=10) | IW-1973 40 mg QD/QD (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Injection site haemorrhage (General disorders) | 3 | 0 | 1
Injection site injury (General disorders) | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 3
Pseudohypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 3
Dizziness (Nervous system disorders) | 1 | 1 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may publish or disclose the results of the study 24 months after final data lock provided that sponsor can review the publication prior to public release, sponsor can request removal of confidential information of sponsor (not including results of trial), and sponsor can request a publication delay in order to protect potentially patentable information. Furthermore, if a publication committee is developing an initial publication, PI is to delay disclosure until that publication is published.

DOCUMENTS (2):
  • Study Protocol (2017-03-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT03091920/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT03091920/SAP_001.pdf